CLINICAL TRIAL: NCT02045862
Title: A Randomized, Double-Blind, Parallel-Group, Active-Controlled, Multi-center Study to Evaluate the Long-Term Safety and Efficacy of Combination of Solifenacin Succinate With Mirabegron Compared to Solifenacin Succinate and Mirabegron Monotherapy in Subjects With Overactive Bladder
Brief Title: A Multinational Study Comparing the Long-term Efficacy and Safety of Two Medicines, Solifenacin Succinate and Mirabegron Taken Together, or Separately, in Subjects With Symptoms of Overactive Bladder
Acronym: SYNERGY II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 178-CL-102; 2012-005736-29 (EudraCT Number)
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder Overactive; Overactive Bladder; Urgency Incontinence; Urinary Bladder Diseases\Urologic Diseases
Keywords: Solifenacin Succinate; Mirabegron; Urinary Incontinence; Combination Therapy; Urgency; Nocturia; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Nocturia | interventions — Solifenacin Succinate; mirabegron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mirabegron 50 mg (Active Comparator): Participants received mirabegron 50 mg once a day for 52 weeks.
  Interventions: Drug: Mirabegron; Drug: Placebo to match solifenacin
- Solifenacin 5 mg (Active Comparator): Participants received solifenacin 5 mg once a day for 52 weeks.
  Interventions: Drug: Solifenacin succinate; Drug: Placebo to match mirabegron
- Solifenacin 5 mg + Mirabegron 50 mg (Experimental): Participants received solifenacin 5 mg and mirabegron 50 mg once a day for 52 weeks.
  Interventions: Drug: Solifenacin succinate; Drug: Mirabegron

INTERVENTIONS:
Drug: Solifenacin succinate — Participants received solifenacin 5 mg orally once a day at the same time each day.
  Other Names: Vesicare; Vesitrim; YM905; Vesikur
  Arms: Solifenacin 5 mg; Solifenacin 5 mg + Mirabegron 50 mg
Drug: Mirabegron — Participants received mirabegron 50 mg orally once a day at the same time each day.
  Other Names: Myrbetriq; YM178; Betmiga; Betanis
  Arms: Mirabegron 50 mg; Solifenacin 5 mg + Mirabegron 50 mg
Drug: Placebo to match solifenacin — Participants received placebo to match solifenacin 5 mg orally once a day at the same time each day. This intervention was given to maintain the blind during the study.
  Arms: Mirabegron 50 mg
Drug: Placebo to match mirabegron — Participants received placebo to match mirabegron 50 mg orally once a day at the same time each day. This intervention was given to maintain the blind during the study.
  Arms: Solifenacin 5 mg

SUMMARY:
The purpose of this study was to examine how well the combination of two medicines (solifenacin succinate and mirabegron) worked compared to each medicine alone in the treatment of bladder problems, and how safe they were for long term use.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion at Screening (Visit 1):

* Subject had completed study 178-CL-101 or study 905-EC-012 (This inclusion criterion would no longer apply once the recruitment for study 178-CL-101 and study 905-EC-012 had been completed. In that case the subject had to have symptoms of "wet" OAB (urinary frequency and urgency with incontinence) for at least 3 months);
* Subject was willing and able to complete the micturition diary and questionnaires correctly and able to measure his/her vital signs at home at stipulated time points, using the device provided by the study personnel, and to adequately record the readings;

Main Inclusion at Randomization (Visit 2):

* Subject had a micturition frequency of on average ≥ 8 times per 24-hour period during the last 7 days of the micturition diary period (incontinence episode should not be counted as a micturition).
* Subject had experienced at least 3 incontinence episodes during the last 7 days of the micturition diary period.
* Subject had experienced on average at least 1 urgency episode (grade 3 or 4 on Patient Perception of Intensity of Urgency Scale [PPIUS]) per 24-hour period during the 7-day micturition diary period.

Exclusion Criteria:

Main Exclusion at Screening (Visit 1):

* Subject had clinically significant bladder outflow obstruction at risk of urinary retention;
* Subject had significant PVR volume (> 150 mL);
* Subject had significant stress incontinence or mixed stress/urgency incontinence where stress is the predominant factor;
* Subject has an indwelling catheter or practices intermittent self-catheterization;
* Subject had evidence of a UTI (urine culture containing > 100,000 cfu/mL), chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs;
* Subject had intravesical treatment in the past 12 months with e.g., botulinum toxin, resiniferatoxin, capsaicin;

Main Exclusion at Randomization (Visit 2):

* Subject had evidence of a urinary tract infection (UTI) (urine culture containing > 100,000 cfu/mL) as assessed in the Screening visit (V1) samples. The subject could be rescreened after successful treatment of the UTI (confirmed by a dipstick negative for nitrite).
* Subject had an average total daily urine volume > 3000 mL as recorded in the micturition diary period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1829 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2016-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (251):
- United States (75):
  - Site US10049, Mobile, Alabama
  - Site US10112, Mobile, Alabama
  - Site US10104, Chandler, Arizona
  - Site US10021, Phoenix, Arizona
  - Site US10122, Anaheim, California
  - Site US10082, Hawaiian Gardens, California
  - Site US10132, Los Angeles, California
  - Site US10133, Los Angeles, California
  - Site US10149, Paramount, California
  - Site US10003, San Diego, California
  - Site US10106, Tarzana, California
  - Site US10595, Valley Village, California
  - Site US10053, Wheat Ridge, Colorado
  - Site US10060, Bradenton, Florida
  - Site US10097, Hialeah, Florida
  - Site US10148, Hialeah, Florida
  - Site US10153, Hialeah, Florida
  - Site US10091, Jupiter, Florida
  - Site US10150, New Port Richey, Florida
  - Site US10124, Orlando, Florida
  - Site US10134, Orlando, Florida
  - Site US10009, Pembroke Pines, Florida
  - Site US10554, Plantation, Florida
  - Site US10037, Alpharetta, Georgia
  - Site US10127, Roswell, Georgia
  - Site US10120, Sandy Springs, Georgia
  - Site US10078, Wichita, Kansas
  - Site US10088, Lake Charles, Louisiana
  - Site US10025, Shreveport, Louisiana
  - Site US10558, Hanover, Maryland
  - Site US10282, Boston, Massachusetts
  - Site US10114, Watertown, Massachusetts
  - Site US10110, Billings, Montana
  - Site US10154, Missoula, Montana
  - Site US10553, Lincoln, Nebraska
  - Site US10002, Englewood, New Jersey
  - Site US10047, Lawrenceville, New Jersey
  - Site US10011, Albuquerque, New Mexico
  - Site US10015, Albuquerque, New Mexico
  - Site US10026, Garden City, New York
  - Site US10040, Kingston, New York
  - Site US10168, New York, New York
  - Site US10126, Newburgh, New York
  - Site US10028, Poughkeepsie, New York
  - Site US10076, Concord, North Carolina
  - Site US10129, Raleigh, North Carolina
  - Site US10062, Winston-Salem, North Carolina
  - Site US10050, Cleveland, Ohio
  - Site US10067, Wadsworth, Ohio
  - Site US10109, Oklahoma City, Oklahoma
  - Site US10541, Medford, Oregon
  - Site US10008, Bala-Cynwyd, Pennsylvania
  - Site US10017, Philadelphia, Pennsylvania
  - Site US10167, Pittsburgh, Pennsylvania
  - Site US10250, Pittsburgh, Pennsylvania
  - Site US10248, Pittsburgh, Pennsylvania
  - Site US10063, Uniontown, Pennsylvania
  - Site US10012, West Reading, Pennsylvania
  - Site US10166, Charleston, South Carolina
  - Site US10079, Mt. Pleasant, South Carolina
  - Site US10023, Simpsonville, South Carolina
  - Site US10101, Summerville, South Carolina
  - Site US10006, Kingsport, Tennessee
  - Site US10065, Corpus Christi, Texas
  - Site US10085, Houston, Texas
  - Site US10219, Houston, Texas
  - Site US10093, Houston, Texas
  - Site US10090, Hurst, Texas
  - Site US10105, San Antonio, Texas
  - Site US10111, San Antonio, Texas
  - Site US10083, Virginia Beach, Virginia
  - Site US10013, Burien, Washington
  - Site US10004, Mountlake Terrace, Washington
  - Site US10155, Seattle, Washington
  - Site US10135, Walla Walla, Washington
- Australia (11):
  - Site AU61005, Broadmeadow, New South Wales
  - Site AU61007, Randwick, New South Wales
  - Site AU61021, Randwick, New South Wales
  - Site AU61011, Wollongong, New South Wales
  - Site AU61022, Brisbane, Queensland
  - Site AU61010, Nambour, Queensland
  - Site AU61019, Sherwood, Queensland
  - Site AU61015, Daw Park, South Australia
  - Site AU61025, Footscray, Victoria
  - Site AU61002, Parkville, Victoria
  - Site AU61004, Perth, Western Australia
- Belgium (3):
  - Site BE32004, Ghent
  - Site BE32014, Roeselare
  - Site BE32012, Sint-Truiden
- Bulgaria (4):
  - Site BG35908, Plovdiv
  - Site BG35902, Rousse
  - Site BG35905, Sofia
  - Site BG35903, Sofia
- Canada (15):
  - Site CA15035, Edmonton, Alberta
  - Site CA15033, Vancouver, British Columbia
  - Site CA15008, Saint John, New Brunswick
  - Site CA15001, Barrie, Ontario
  - Site CA15006, Brampton, Ontario
  - Site CA15003, Brantford, Ontario
  - Site CA15007, Kitchener, Ontario
  - Site CA15013, Toronto, Ontario
  - Site CA15004, Toronto, Ontario
  - Site CA15026, Drummondville, Quebec
  - Site CA15039, Lévis, Quebec
  - Site CA15020, Montreal, Quebec
  - Site CA15025, Québec, Quebec
  - Site CA15027, Sherbrooke, Quebec
  - Site CA15040, Montreal
- Czechia (11):
  - Site CZ42015, Brno
  - Site CZ42003, Hradec Králové
  - Site CZ42001, Hradec Králové
  - Site CZ42010, Olomouc
  - Site CZ42014, Ostrava
  - Site CZ42005, Pilsen
  - Site CZ42008, Prague
  - Site CZ42007, Prague
  - Site CZ42013, Sternberk
  - Site CZ42009, Uherské Hradiště
  - Site CZ42006, Ústí nad Labem
- Site DK45013, Aarhus, Denmark
- Site EE37201, Pärnu, Estonia
- Site FI35801, Kouvola, Finland
- Germany (12):
  - Site DE49034, Munich, Bavaria
  - Site DE49032, Duisburg, North Rhine-Westphalia
  - Site DE49031, Bergisch Gladbach, Northwest
  - Site DE49013, Leipzig, Saxony
  - Site DE49003, Eisleben Lutherstadt, Saxony-Anhalt
  - Site DE49008, Bad Ems
  - Site DE49002, Duisburg
  - Site DE49010, Ganderkesee
  - Site DE49011, Halle
  - Site DE49001, Neustadt in Sachsen
  - Site DE49026, Rostock
  - Site DE49014, Sangerhausen
- Hungary (6):
  - Site HU36007, Kecskemét, Bacs-Kiskun Megye
  - Site HU36005, Pécs, Baranya
  - Site HU36003, Csongrád, Csongrád megye
  - Site HU36001, Szentes, Csongrád megye
  - Site HU36013, Sopron, Győr-Moson-Sopron
  - Site HU36012, Veszprém, Veszprém megye
- Italy (4):
  - Site IT39022, Ancona
  - Site IT39007, Avellino
  - Site IT39001, Latina
  - Site IT39020, Milan
- Latvia (3):
  - Site LV37102, Liepāja
  - Site LV37103, Olaine
  - Site LV37105, Riga
- Lithuania (8):
  - Site LT37008, Kaunas
  - Site LT37004, Kaunas
  - Site LT37011, Kaunas
  - Site LT37012, Klaipėda
  - Site LT37010, Vilnius
  - Site LT37003, Vilnius
  - Site LT37007, Vilnius
  - Site LT37009, Vilnius
- Site MY60002, Petaling Jaya, Malaysia
- Site MX52003, Mexico City, Mexico City, Mexico
- Netherlands (4):
  - Site NL31006, Enschede, NL
  - Site NL31002, Amsterdam
  - Site NL31005, Nijmegen
  - Site NL31010, Sneek
- New Zealand (4):
  - Site NZ64001, Christchurch, Canterbury
  - Site NZ64002, Nelson
  - Site NZ64003, Tauranga
  - Site NZ64006, Whangarei
- Norway (3):
  - Site NO47007, Ålesund
  - Site NO47006, Hamar
  - Site NO47008, Lierskogen
- Poland (12):
  - Site PL48018, Bialystok
  - Site PL48013, Chorzów
  - Site PL48014, Gdynia
  - Site PL48004, Lodz
  - Site PL48010, Lublin
  - Site PL48011, Mysłowice
  - Site PL48016, Opole
  - Site PL48005, Piaseczno
  - Site PL48012, Warsaw
  - Site PL48003, Warsaw
  - Site PL48001, Warsaw
  - Site PL48019, Wroclaw
- Romania (6):
  - Site RO40014, Cluj-Napoca, Cluj
  - Site RO40004, Bucharest
  - Site RO40001, Bucharest
  - Site RO40005, Bucharest
  - Site RO40010, Sibiu
  - Site RO40002, Timișoara
- Russia (7):
  - Site RU70015, Kazan'
  - Site RU70023, Penza
  - Site RU70019, Saint Petersburg
  - Site RU70002, Saint Petersburg
  - Site RU70022, Saint Petersburg
  - Site RU70014, Saint Petersburg
  - Site RU70018, Ufa
- Singapore (2):
  - Site SG65002, Singapore
  - Site SG65003, Singapore
- Slovakia (8):
  - Site SK42105, Bratislava
  - Site SK42107, Košice
  - Site SK42101, Košice
  - Site SK42103, Nitra
  - Site SK42108, Poprad
  - Site SK42104, Prešov
  - Site SK42102, Trenčín
  - Site SK42106, Trenčín
- Site SI38604, Murska Sobota, Slovenia
- South Africa (5):
  - Site ZA27001, Centurion, Gauteng
  - Site ZA27002, Roodepoort, Gauteng
  - Site ZA27006, Durban, KwaZulu-Natal
  - Site ZA27013, Meyerspark, Pretoria
  - Site ZA27007, Paarl, Western Cape
- South Korea (20):
  - Site KR82004, Suwon, Gyeonggi-do
  - Site KR82014, Bucheon-si, Gyunggido
  - Site KR82012, Seoul, Gyunggido
  - Site KR82010, Jeonju, Jeollabuk-do South Korea
  - Site KR82006, Busan
  - Site KR82016, Busan
  - Site KR82005, Daegu
  - Site KR82029, Daegu
  - Site KR82019, Daejeon
  - Site KR82023, Incheon
  - Site KR82003, Seoul
  - Site KR82021, Seoul
  - Site KR82020, Seoul
  - Site KR82030, Seoul
  - Site KR82013, Seoul
  - Site KR82017, Seoul
  - Site KR82002, Seoul
  - Site KR82008, Seoul
  - Site KR82015, Seoul
  - Site KR82001, Seoul
- Spain (4):
  - Site ES34004, Madrid
  - Site ES34015, Madrid
  - Site ES34009, Madrid
  - Site ES34002, Valencia
- Sweden (6):
  - Site SE46007, Borås
  - Site SE46005, Malmo
  - Site SE46016, Stockholm
  - Site SE46012, Stockholm
  - Site SE46003, Stockholm
  - Site SE46009, Uppsala
- Thailand (2):
  - Site TH66008, Bangkok
  - Site TH66009, Khon Kaen
- Ukraine (7):
  - Site UA38002, Cherenigiv
  - Site UA38015, Chernivtsi
  - Site UA38013, Dnipro
  - Site UA38007, Kiev
  - Site UA38003, Kyiv
  - Site UA38010, Kyiv
  - Site UA38008, Zaporizhzhya
- United Kingdom (3):
  - Site GB44001, Sheffield, South Yorkshire
  - Site GB44006, Plymouth
  - Site GB44009, Watford

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Gratzke C, van Maanen R, Chapple C, Abrams P, Herschorn S, Robinson D, Ridder A, Stoelzel M, Paireddy A, Yoon SJ, Al-Shukri S, Rechberger T, Mueller ER. Long-term Safety and Efficacy of Mirabegron and Solifenacin in Combination Compared with Monotherapy in Patients with Overactive Bladder: A Randomised, Multicentre Phase 3 Study (SYNERGY II). Eur Urol. 2018 Oct;74(4):501-509. doi: 10.1016/j.eururo.2018.05.005. Epub 2018 Jun 1. PMID 29866467
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=246

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had symptoms of "wet" overactive bladder (OAB) (urgency, urinary frequency and urgency incontinence) for ≥ 3 months were enrolled in 251 centers globally. A majority of the participants were recruited from participants who enrolled and completed studies 178-CL-101 (NCT01972841) or 905-EC-012 (NCT01908829).
Pre-assignment Details: A total of 2084 participants were screened, 2063 participants received placebo run-in treatment and 1829 participants were randomized into 1 of 3 treatment arms in a 1:1:4 ratio in the 52-week double-blind treatment period. Randomization was stratified by sex, age group (< 65 years, ≥ 65 years) and geographic region.
Period: Overall Study
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Started | 306 | 305 | 1218
Treated | 306 | 303 | 1210
Completed | 267 | 265 | 1092
Not Completed | 39 | 40 | 126
Not completed — Death | 0 | 0 | 1
Not completed — Miscellaneous | 5 | 0 | 8
Not completed — Withdrawal by Patient | 18 | 27 | 57
Not completed — Protocol Violation | 0 | 0 | 6
Not completed — Lack of Efficacy | 8 | 4 | 13
Not completed — Randomized but not Received Study Drug | 0 | 2 | 8
Not completed — Adverse Event | 7 | 5 | 27
Not completed — Lost to Follow-up | 1 | 2 | 6

BASELINE CHARACTERISTICS:
Population: The analysis population was the randomized analysis set (RAS), which comprised of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg | Total
Number analyzed (Participants) | 306 | 305 | 1218 | 1829
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (12.7) | 59.0 (13.3) | 58.3 (13.0) | 58.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 243 | 245 | 973 | 1461
  Male | 63 | 60 | 245 | 368
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 266 | 265 | 1066 | 1597
  Black or African American | 5 | 4 | 27 | 36
  Asian | 31 | 33 | 119 | 183
  Other | 4 | 3 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 54 | 84
  Not Hispanic or Latino | 291 | 290 | 1164 | 1745
Mean Number of Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: incontinence episodes/24 hours] — An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to the first dose of double-blind treatment. Population: Full analysis set (FAS), which consisted of all randomized participants who took ≥ 1 dose of double-blind treatment, reported ≥ 1 micturition in the baseline diary and ≥ 1 micturition postbaseline, reported ≥ 1 incontinence episode in the baseline diary and excluded participants from 2 sites due to protocol noncompliance and data integrity issues.
  incontinence episodes/24 hours
    number analyzed (Participants) | 302 | 299 | 1193 | 1794
    (all) | 3.15 (3.56) | 3.10 (3.58) | 3.04 (3.17) | 3.07 (3.31)
Mean Number of Micturitions per 24 Hours [Mean (Standard Deviation); unit: micturitions/24 hours] — A micturition was defined as any voluntary act of passing urine (excluding incontinence only episodes). The mean number of micturitions per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to the first dose of double-blind treatment. Population: FAS population
  micturitions/24 hours
    number analyzed (Participants) | 302 | 299 | 1193 | 1794
    (all) | 10.51 (2.41) | 10.76 (2.83) | 10.55 (2.73) | 10.58 (2.70)
Mean Volume Voided per Micturition [Mean (Standard Deviation); unit: mL] — The mean volume voided per micturition was calculated from the data recorded by the participant during 3 consecutive days with volume measurements during the 7-day micturition diary period prior to first dose of double-blind treatment. Population: FAS population with available data at baseline
  mL
    number analyzed (Participants) | 302 | 299 | 1190 | 1791
    (all) | 161.00 (60.16) | 160.70 (58.49) | 159.29 (58.40) | 159.82 (58.69)
Number of Incontinence Episodes per Week [Mean (Standard Deviation); unit: incontinence episodes/week] — An incontinence episode was defined as the complaint of any involuntary leakage of urine. The number of incontinence episodes per week was the total number of times a participant recorded an incontinence episode in a micturition diary for 7 days prior to the first dose of double-blind treatment. Population: FAS population
  incontinence episodes/week
    number analyzed (Participants) | 302 | 299 | 1193 | 1794
    (all) | 21.8 (24.8) | 21.6 (25.0) | 20.9 (21.9) | 21.2 (22.9)
Mean Number of Urgency Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: urgency incontinence episodes/24 hours] — An urgency incontinence episode was defined as the involuntary leakage of urine accompanied by or immediately preceded by urgency. The mean number of urgency incontinence episodes per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to the first dose of double-blind treatment. Population: FAS population with ≥ 1 urgency incontinence episode at baseline
  urgency incontinence episodes/24 hours
    number analyzed (Participants) | 302 | 297 | 1187 | 1786
    (all) | 2.86 (3.29) | 2.91 (3.49) | 2.74 (2.78) | 2.79 (3.00)
Number of Urgency Incontinence Episodes per Week [Mean (Standard Deviation); unit: urgency incontinence episodes/week] — An urgency incontinence episode was defined as the involuntary leakage of urine accompanied by or immediately preceded by urgency. The number of urgency incontinence episodes per week was the total number of times a participant recorded an urgency incontinence episode in a micturition diary for 7 days prior to the first dose of double-blind treatment. Population: FAS population with ≥ 1 urgency incontinence episode at baseline
  urgency incontinence episodes/week
    number analyzed (Participants) | 302 | 297 | 1187 | 1786
    (all) | 19.8 (22.8) | 20.2 (24.5) | 18.9 (19.1) | 19.3 (20.7)
Mean Number of Urgency Episodes (Grade 3 or 4) per 24 Hours [Mean (Standard Deviation); unit: urgency episodes/24 hours] — Urgency was defined as a complaint of a sudden, compelling desire to pass urine, which is difficult to defer. An urgency episode was defined as any micturition or incontinence episode recorded by the participant in a micturition diary for 7 days prior to the first dose of double-blind treatment as 3 or 4 on the Patient Perception of Intensity of Urgency Scale (PPIUS), where 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could delay voiding a short while; 3 = Severe urgency, could not delay voiding; 4 = Urge incontinence, leaked before arriving to the toilet. Population: FAS population with ≥ 1 urgency episode at baseline
  urgency episodes/24 hours
    number analyzed (Participants) | 302 | 299 | 1193 | 1794
    (all) | 6.34 (4.16) | 6.63 (4.08) | 6.53 (3.69) | 6.51 (3.84)
Mean Number of Nocturia Episodes per 24 Hours [Mean (Standard Deviation); unit: nocturia episodes/24 hours] — A nocturia episode was defined as waking at night 1 or more times to void (i.e., any voiding associated with sleep disturbance between the time the participant goes to bed with the intention to sleep until the time the participant gets up in the morning with the intention to stay awake). The mean number of nocturia episodes per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to the first dose of double-blind treatment. Population: FAS population with ≥ 1 nocturia episode at baseline
  nocturia episodes/24 hours
    number analyzed (Participants) | 262 | 252 | 1027 | 1541
    (all) | 1.48 (0.95) | 1.58 (0.94) | 1.49 (0.94) | 1.51 (0.94)
Number of Nocturia Episodes per Week [Mean (Standard Deviation); unit: nocturia episodes/week] — A nocturia episode was defined as waking at night 1 or more times to void (i.e., any voiding associated with sleep disturbance between the time the participant goes to bed with the intention to sleep until the time the participant gets up in the morning with the intention to stay awake). The number of nocturia episodes per week was the number of times a participant recorded a nocturia episode in a micturition diary for 7 days prior to the first dose of double-blind treatment. Population: FAS population with ≥ 1 nocturia episode at baseline
  nocturia episodes/week
    number analyzed (Participants) | 262 | 252 | 1027 | 1541
    (all) | 10.3 (6.6) | 11.0 (6.6) | 10.4 (6.5) | 10.4 (6.5)
Mean Number of Pads Used per 24 Hours [Mean (Standard Deviation); unit: pads/24 hours] — The mean number of pads used per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to the first dose of double-blind treatment. Population: FAS population with ≥ 1 pad used at baseline
  pads/24 hours
    number analyzed (Participants) | 201 | 193 | 771 | 1165
    (all) | 2.51 (3.76) | 2.77 (3.15) | 2.58 (2.59) | 2.60 (2.91)
Number of Pads Used per Week [Mean (Standard Deviation); unit: pads/week] — The number of pads used per week was the number of times a participant recorded a new pad used during the 7-day micturition diary period prior to the first dose of double-blind treatment. Population: FAS population with ≥ 1 pad used at baseline
  pads/week
    number analyzed (Participants) | 201 | 193 | 771 | 1165
    (all) | 17.3 (26.1) | 19.2 (22.0) | 17.7 (17.6) | 17.9 (20.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) observed after taking the first dose of double-blind treatment until 14 days after taking the last dose of double-blind treatment for non-serious AEs and until 30 days after taking the last dose of double-blind treatment for serious adverse events (SAEs). This included abnormal laboratory tests, vital signs or electrocardiogram data that were defined as AEs if the abnormality induced clinical signs or symptoms, required active intervention, interruption or discontinuation of study drug or was clinically significant in the investigator's opinion. The severity of each AE was defined according to the following: Mild (No disruption of normal daily activities); Moderate (Affected normal daily activities) and Severe (Inability to perform daily activities).
Time Frame: From first dose of double-blind study drug up to 30 days after last dose of double-blind study drug (up to 56 weeks)
Population: The analysis population was the safety analysis set (SAF), which consisted of all participants who received ≥ 1 dose of double-blind study drug and excluded participants from one site due to protocol noncompliance.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 305 | 303 | 1206
Participants
  Any TEAEs | 126 | 134 | 596
  Mild TEAEs | 61 | 69 | 306
  Moderate TEAEs | 52 | 58 | 238
  Severe TEAEs | 13 | 7 | 52
  Drug-related TEAEs | 35 | 42 | 200
  Serious TEAEs | 8 | 8 | 51
  Drug-related Serious TEAEs | 1 | 0 | 0
  TEAEs Leading to Discontuation of Study Drug | 7 | 5 | 25
  Drug-related TEAEs Leading to Discont. of Drug | 4 | 4 | 17
  TEAEs Leading to Death | 0 | 0 | 1

2. Primary Outcome: Change From Baseline to End of Treatment (EoT) in Mean Number of Incontinence Episodes Per 24 Hours
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to the baseline and week 52 clinic visits.
Time Frame: Baseline and Week 52
Population: FAS population; Last observation carried forward (LOCF) was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 301 | 297 | 1184
incontinence episodes | -1.58 (0.11) | -1.90 (0.11) | -2.03 (0.05)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference vs. Mirabegron 50 mg: Difference of the adjusted mean (i.e., least squares mean) was calculated by subtracting the adjusted mean of the mirabegron monotherapy group from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p < 0.001, Stratified Rank ANCOVA — The 2-sided P value was for pairwise comparisons between the combination therapy group and the corresponding monotherapy group from the stratified rank ANCOVA; Least Squares Mean Difference = -0.45, 95% CI 2-sided [-0.69 to -0.21], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference vs. Solifenacin 5 mg: Difference of the adjusted mean (i.e., least squares mean) was calculated by subtracting the adjusted mean of the solifenacin monotherapy group from the adjusted mean of the combination group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.002, Stratified Rank ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.13, 95% CI 2-sided [-0.37 to 0.11], Standard Error of Mean 0.12

3. Primary Outcome: Change From Baseline to EoT in Mean Number of Micturitions Per 24 Hours
Description: A micturition was defined as any voluntary urination (excluding incontinence only episodes). The mean number of micturitions per 24 hours was calculated from data recorded by the participant in a micturition diary for 7-days before the baseline and week 52 clinic visits.
Time Frame: Baseline and Week 52
Population: FAS population; LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 301 | 297 | 1184
micturitions | -2.10 (0.13) | -2.16 (0.13) | -2.58 (0.07)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — The 2-sided P value was for pairwise comparisons between the combination therapy group and the corresponding monotherapy group from the ANCOVA model; Least Squares Mean Difference = -0.48, 95% CI 2-sided [-0.77 to -0.20], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.004, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean Difference = -0.42, 95% CI 2-sided [-0.71 to -0.13], Standard Error of Mean 0.15

4. Secondary Outcome: Change From Baseline to EoT in Mean Volume Voided Per Micturition
Description: The mean volume voided per micturition was calculated from the data recorded by the participant during 3 consecutive days with volume measurements during the 7-day micturition diary period.
Time Frame: Baseline and Week 52
Population: FAS population with baseline and at least one post-baseline measurement; LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 289 | 293 | 1162
mL | 21.83 (3.12) | 24.90 (3.10) | 37.67 (1.55)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = 15.84, 95% CI 2-sided [8.99 to 22.69], Standard Error of Mean 3.49
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = 12.77, 95% CI 2-sided [5.98 to 19.57], Standard Error of Mean 3.47

5. Secondary Outcome: Change From Baseline to EoT in Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score
Description: The OAB-q is a self-reported questionnaire with items relating to symptom bother and health-related quality of life (HRQoL). The symptom bother portion consists of 8 items, rated on a 6-point Likert scale (1 through 6). The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 (least severity) to 100 (worst severity). A negative change from baseline indicated an improvement.
Time Frame: Baseline and Week 52
Population: FAS population with baseline and at least one post-baseline measurement; LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 290 | 294 | 1163
units on a scale | -21.96 (1.14) | -24.91 (1.13) | -29.51 (0.57)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -7.55, 95% CI 2-sided [-10.05 to -5.05], Standard Error of Mean 1.27
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -4.60, 95% CI 2-sided [-7.09 to -2.12], Standard Error of Mean 1.27

6. Secondary Outcome: Change From Baseline to EoT in the Patient's Assessment of Treatment Satisfaction-Visual Analogue Scale (TS-VAS)
Description: The TS-VAS is a visual analogue scale which asks participants to rate their satisfaction with the treatment by placing a vertical mark on a line that runs from 0 (No, not at all) on the left to 10 (Yes, completely) on the right. A positive change from baseline indicated improvement.
Time Frame: Baseline and Week 52
Population: FAS population with baseline and at least one post-baseline measurement; LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 289 | 294 | 1163
units on a scale | 2.19 (0.12) | 2.15 (0.12) | 2.73 (0.06)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = 0.55, 95% CI 2-sided [0.28 to 0.82], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = 0.59, 95% CI 2-sided [0.32 to 0.86], Standard Error of Mean 0.14

7. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9 and 12 in Mean Number of Incontinence Episodes Per 24 Hours
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to the baseline and prior to each visit.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
incontinence episodes
  Month 1: number analyzed (Participants) | 291 | 288 | 1158
  Month 1 | -0.97 (0.10) | -1.29 (0.11) | -1.45 (0.05)
  Month 3: number analyzed (Participants) | 282 | 288 | 1137
  Month 3 | -1.31 (0.11) | -1.71 (0.11) | -1.78 (0.05)
  Month 6: number analyzed (Participants) | 266 | 273 | 1107
  Month 6 | -1.42 (0.11) | -1.78 (0.11) | -1.93 (0.05)
  Month 9: number analyzed (Participants) | 264 | 261 | 1070
  Month 9 | -1.53 (0.11) | -1.90 (0.11) | -2.00 (0.06)
  Month 12: number analyzed (Participants) | 258 | 256 | 1048
  Month 12 | -1.67 (0.11) | -1.92 (0.11) | -2.06 (0.06)

8. Secondary Outcome: Number of Incontinence Episodes During the 7-Day Micturition Diary Period Prior to Each Visit
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The number of incontinence episodes was the total number of times a participant records an incontinence episode during the 7-day micturition diary period prior to each visit.
Time Frame: Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point; LOCF was used for EoT.
Measure: Mean (Standard Error); unit: incontinence episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
incontinence episodes
  Month 1: number analyzed (Participants) | 291 | 288 | 1158
  Month 1 | 14.88 (1.52) | 12.41 (1.22) | 10.80 (0.58)
  Month 3: number analyzed (Participants) | 282 | 288 | 1137
  Month 3 | 12.23 (1.12) | 9.23 (1.02) | 8.33 (0.52)
  Month 6: number analyzed (Participants) | 266 | 273 | 1107
  Month 6 | 10.62 (1.08) | 8.18 (1.01) | 7.28 (0.48)
  Month 9: number analyzed (Participants) | 264 | 261 | 1070
  Month 9 | 10.53 (1.19) | 7.28 (0.91) | 6.74 (0.45)
  Month 12: number analyzed (Participants) | 258 | 256 | 1048
  Month 12 | 9.09 (1.10) | 7.06 (0.94) | 6.10 (0.46)
  EoT: number analyzed (Participants) | 301 | 297 | 1184
  EoT | 10.32 (1.08) | 8.09 (0.94) | 6.85 (0.47)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Rate ratio of number of incontinence episodes during the EoT 7-day diary between the combination therapy group and the mirabegron monotherapy group was calculated from a negative binomial regression model incl. treatment group, sex, age group (< 65, ≥ 65 years), geographic region and previous study history as factors, log(number of incontinence episodes divided by number of valid diary days) at baseline included as a covariate and number of valid diary day at EoT as the offset variable; Test type: Superiority; p < 0.001, Mixed Effects Poisson-Negative Binomial; Rate Ratio = 0.67, 95% CI 2-sided [0.54 to 0.84], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Rate ratio of number of incontinence episodes during the EoT 7-day diary between the combination therapy group and the solifenacin monotherapy group was calculated from a negative binomial regression model incl. treatment group, sex, age group (< 65, ≥ 65 years), geographic region and previous study history as factors, log(number of incontinence episodes divided by number of valid diary days) at baseline included as a covariate and number of valid diary day at EoT as the offset variable; Test type: Superiority; p = 0.029, Mixed Effects Poisson-Negative Binomial; Rate Ratio = 0.77, 95% CI 2-sided [0.61 to 0.97], Standard Error of Mean 0.12

9. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in Number of Incontinence Episodes During the 7-Day Micturition Diary Period Prior to Each Visit
Description: as for outcome 8
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point; LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
incontinence episodes
  Month 1: number analyzed (Participants) | 291 | 288 | 1158
  Month 1 | -6.77 (0.73) | -9.17 (0.73) | -10.31 (0.36)
  Month 3: number analyzed (Participants) | 282 | 288 | 1137
  Month 3 | -9.21 (0.76) | -12.05 (0.75) | -12.55 (0.38)
  Month 6: number analyzed (Participants) | 266 | 273 | 1107
  Month 6 | -10.36 (0.76) | -12.50 (0.75) | -13.49 (0.37)
  Month 9: number analyzed (Participants) | 264 | 261 | 1070
  Month 9 | -10.62 (0.76) | -13.51 (0.77) | -14.06 (0.38)
  Month 12: number analyzed (Participants) | 258 | 256 | 1048
  Month 12 | -11.84 (0.77) | -13.47 (0.77) | -14.43 (0.38)
  EoT: number analyzed (Participants) | 301 | 297 | 1184
  EoT | -11.17 (0.75) | -13.37 (0.75) | -14.29 (0.37)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference vs. Mirabegron 50 mg (EoT): Difference of the adjusted mean is calculated by subtracting the adjusted mean of the mirabegron monotherapy group from the adjusted mean of the combination therapy group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p < 0.001, Stratified Rank ANCOVA — The two-sided p-value is for pairwise comparisons between the combination therapy group and the mirabegron monotherapy group from stratified rank ANCOVA; Least Squares Mean Difference = -3.12, 95% CI 2-sided [-4.76 to -1.49], Standard Error of Mean 0.83
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference vs. Solifenacin 5 mg (EoT): Difference of the adjusted mean is calculated by subtracting the adjusted mean of the solifenacin monotherapy group from the adjusted mean of the combination therapy group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p < 0.001, Stratified Rank ANCOVA — The two-sided p-value is for pairwise comparisons between the combination therapy group and the solifenacin monotherapy group from stratified rank ANCOVA; Least Squares Mean Difference = -0.93, 95% CI 2-sided [-2.57 to 0.72], Standard Error of Mean 0.84

10. Secondary Outcome: Number of Incontinence-Free Days During the 7-Day Micturition Diary Period Prior to Each Visit
Description: The number of incontinence-free days was the number of valid diary days during the 7-day micturition diary period prior to each visit with no incontinence episodes recorded.
Time Frame: Months 1, 3, 6, 9, 12
Population: FAS population with with data available at each time point; LOCF was used for EoT.
Measure: Mean (Standard Error); unit: incontinence-free days
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
incontinence-free days
  Month 1: number analyzed (Participants) | 291 | 288 | 1158
  Month 1 | 2.73 (0.15) | 3.35 (0.17) | 3.46 (0.08)
  Month 3: number analyzed (Participants) | 282 | 288 | 1137
  Month 3 | 3.30 (0.17) | 3.98 (0.17) | 4.17 (0.08)
  Month 6: number analyzed (Participants) | 266 | 273 | 1107
  Month 6 | 3.64 (0.17) | 4.08 (0.17) | 4.44 (0.08)
  Month 9: number analyzed (Participants) | 264 | 261 | 1070
  Month 9 | 3.97 (0.18) | 4.33 (0.17) | 4.56 (0.08)
  Month 12: number analyzed (Participants) | 258 | 256 | 1048
  Month 12 | 4.23 (0.18) | 4.5 (0.18) | 4.81 (0.08)
  EoT: number analyzed (Participants) | 301 | 297 | 1184
  EoT | 3.98 (0.17) | 4.29 (0.16) | 4.64 (0.08)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio vs. Mirabegron 50 mg (EoT): Odds ratio was from a overdispersed binomial regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and log transformed baseline mean number of incontinence episodes per 24 hours as a covariate; Test type: Superiority; p < 0.001, Overdispersed Binomial Regression; Odds Ratio (OR) = 1.60, 95% CI 2-sided [1.26 to 2.01]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio vs. Solifenacin 5 mg (EoT): Odds ratio was from a overdispersed binomial regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and log transformed baseline mean number of incontinence episodes per 24 hours as a covariate; Test type: Superiority; p = 0.009, Overdispersed Binomial Regression; Odds Ratio (OR) = 1.38, 95% CI 2-sided [1.08 to 1.75]

11. Secondary Outcome: Number of Incontinence-Free Days With < 8 Micturitions Per Day During the 7-Day Micturition Diary Period Prior to Each Visit
Description: The number of incontinence-free days with < 8 micturitions per day was the number of valid diary days during the 7-day micturition diary period with no incontinence episodes recorded and with < 8 micturitions per day.
Time Frame: Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point; LOCF was used for EoT.
Measure: Mean (Standard Error); unit: days
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
days
  Month 1: number analyzed (Participants) | 291 | 288 | 1158
  Month 1 | 1.03 (0.10) | 1.01 (0.10) | 1.33 (0.06)
  Month 3: number analyzed (Participants) | 282 | 288 | 1137
  Month 3 | 1.24 (0.12) | 1.48 (0.13) | 1.91 (0.07)
  Month 6: number analyzed (Participants) | 266 | 273 | 1107
  Month 6 | 1.56 (0.14) | 1.66 (0.14) | 2.13 (0.08)
  Month 9: number analyzed (Participants) | 264 | 261 | 1070
  Month 9 | 1.56 (0.14) | 1.64 (0.14) | 2.20 (0.08)
  Month 12: number analyzed (Participants) | 258 | 256 | 1048
  Month 12 | 1.87 (0.15) | 1.92 (0.15) | 2.54 (0.08)
  EoT: number analyzed (Participants) | 301 | 297 | 1184
  EoT | 1.75 (0.14) | 1.90 (0.14) | 2.43 (0.07)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio vs. Mirabegron 50 mg (EoT): Odds ratio was from a overdispersed binomial regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and log transformed baseline mean number of incontinence episodes per 24 hours and baseline mean number of micturitions per 24 hours as a covariates; Test type: Superiority; p < 0.001, Overdispersed Binomial Regression; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.26 to 2.05]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio vs. Solifenacin 5 mg (EoT): Odds ratio was from a overdispersed binomial regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and log transformed baseline mean number of incontinence episodes per 24 hours and baseline mean number of micturitions per 24 hours as a covariates; Test type: Superiority; p = 0.002, Overdispersed Binomial Regression; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.14 to 1.85]

12. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in Mean Number of Urgency Incontinence Episodes Per 24 Hours
Description: An urgency incontinence episode was defined as the involuntary leakage of urine accompanied by or immediately preceded by urgency. The mean number of urgency incontinence episodes was calculated from data recorded by the participant in a micturition diary for 7 days prior to each visit.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. Only participants with ≥ 1 urgency incontinence episode at baseline were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 297 | 1187
urgency incontinence episodes
  Month 1: number analyzed (Participants) | 291 | 286 | 1152
  Month 1 | -0.93 (0.10) | -1.25 (0.10) | -1.43 (0.05)
  Month 3: number analyzed (Participants) | 282 | 286 | 1132
  Month 3 | -1.30 (0.10) | -1.64 (0.10) | -1.71 (0.05)
  Month 6: number analyzed (Participants) | 266 | 271 | 1101
  Month 6 | -1.40 (0.10) | -1.67 (0.10) | -1.86 (0.05)
  Month 9: number analyzed (Participants) | 264 | 259 | 1066
  Month 9 | -1.60 (0.11) | -1.78 (0.11) | -1.92 (0.05)
  Month 12: number analyzed (Participants) | 258 | 254 | 1043
  Month 12 | -1.60 (0.10) | -1.82 (0.10) | -1.98 (0.05)
  EoT: number analyzed (Participants) | 301 | 295 | 1178
  EoT | -1.51 (0.10) | -1.81 (0.10) | -1.94 (0.05)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference vs. Mirabegron 50 mg (EoT): Difference of the adjusted mean was calculated by subtracting the adjusted mean of the mirabegron monotherapy group from the adjusted mean of the combination therapy group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p < 0.001, Stratified Rank ANCOVA — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -0.43, 95% CI 2-sided [-0.65 to -0.21], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference vs. Solifenacin 5 mg (EoT): Difference of the adjusted mean was calculated by subtracting the adjusted mean of the solifenacin monotherapy group from the adjusted mean of the combination therapy group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.009, Stratified Rank ANCOVA — [p-value comment as in outcome 9, analysis 2]; Least Squares Mean Difference = -0.13, 95% CI 2-sided [-0.36 to 0.09], Standard Error of Mean 0.11

13. Secondary Outcome: Number of Urgency Incontinence Episodes During the 7-Day Micturition Diary Period Prior to Each Visit
Description: An urgency incontinence episode was defined as the involuntary leakage of urine accompanied by or immediately preceeded by urgency. The number of urgency incontinence episodes was the total number of urgency incontinence episodes recorded by the participant during the 7-day micturition diary period prior to each visit.
Time Frame: Months 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 297 | 1187
urgency incontinence episodes
  Month 1: number analyzed (Participants) | 291 | 286 | 1152
  Month 1 | 13.14 (1.42) | 11.21 (1.19) | 8.99 (0.47)
  Month 3: number analyzed (Participants) | 282 | 286 | 1132
  Month 3 | 10.37 (1.00) | 8.12 (0.98) | 6.95 (0.44)
  Month 6: number analyzed (Participants) | 266 | 271 | 1101
  Month 6 | 8.97 (0.95) | 7.31 (0.96) | 5.88 (0.41)
  Month 9: number analyzed (Participants) | 264 | 259 | 1066
  Month 9 | 8.08 (1.01) | 6.51 (0.89) | 5.47 (0.40)
  Month 12: number analyzed (Participants) | 258 | 254 | 1043
  Month 12 | 7.73 (1.00) | 6.06 (0.85) | 4.88 (0.38)
  EoT: number analyzed (Participants) | 301 | 295 | 1178
  EoT | 8.86 (0.98) | 7.04 (0.86) | 5.57 (0.40)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Rate ratio of number of incontinence episodes during the EoT 7-day diary between the combination therapy group and the mirabegron monotherapy group was calculated from a negative binomial regression model incl. treatment group, sex, age group (< 65, ≥65 years), geographic region and previous study history as factors, log(number of urgency incontinence episodes divided by number of valid diary days) included as a covariate and post baseline number of valid diary days at EoT as the offset variable; Test type: Superiority; p < 0.001, Negative Binomial Regression; Rate Ratio = 0.62, 95% CI 2-sided [0.48 to 0.79], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Rate ratio of number of incontinence episodes during the EoT 7-day diary between the combination therapy group and the solifenacin monotherapy group is calculated from a negative binomial regression model incl. treatment group, sex, age group (< 65, ≥ 65 years), geographic region and previous study history as factors, log(number of urgency incontinence episodes divided by number of valid diary days) included as a covariate and post baseline number of valid diary day at EoT as the offset variable; Test type: Superiority; p = 0.023, Negative Binomial Regression; Rate Ratio = 0.75, 95% CI 2-sided [0.58 to 0.96], Standard Error of Mean 0.13

14. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in Number of Urgency Incontinence Episodes During the 7-Day Micturition Diary Period Prior to Each Visit
Description: An urgency incontinence episode was defined as the involuntary leakage of urine accompanied by or immediately preceded by urgency. The number of urgency incontinence episodes was the total number of urgency incontinence episodes recorded by the participant during the 7-day micturition diary period prior to each visit.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
urgency incontinence episodes
  Month 1: number analyzed (Participants) | 291 | 286 | 1152
  Month 1 | -6.45 (0.69) | -8.77 (0.69) | -10.1 (0.34)
  Month 3: number analyzed (Participants) | 282 | 286 | 1132
  Month 3 | -9.06 (0.72) | -11.48 (0.71) | -11.99 (0.36)
  Month 6: number analyzed (Participants) | 266 | 271 | 1101
  Month 6 | -10.09 (0.72) | -11.71 (0.71) | -13.0 (0.35)
  Month 9: number analyzed (Participants) | 264 | 259 | 1066
  Month 9 | -11.1 (0.72) | -12.6 (0.73) | -13.44 (0.36)
  Month 12: number analyzed (Participants) | 258 | 254 | 1043
  Month 12 | -11.27 (0.71) | -12.8 (0.71) | -13.8 (0.35)
  EoT: number analyzed (Participants) | 301 | 295 | 1178
  EoT | -10.61 (0.7) | 12.66 (0.7) | -13.59 (0.35)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.001, Stratified Rank ANCOVA — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -2.98, 95% CI 2-sided [-4.51 to -1.46], Standard Error of Mean 0.78
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference vs. Solifenacin 5 mg (EoT): Difference of the adjusted mean was calculated by subtracting the adjusted mean of the mirabegron monotherapy group from the adjusted mean of the combination therapy group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.006, Stratified Rank ANCOVA — [p-value comment as in outcome 9, analysis 2]; Stratified Rank ANCOVA = -0.93, 95% CI 2-sided [-2.47 to 0.61], Standard Error of Mean 0.78

15. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9 and 12 in Mean Number of Micturitions Per 24 Hours
Description: A micturition was defined as any voluntary urination (excluding incontinence only episodes). The mean number of micturitions per 24 hours was calculated from data recorded by the participant in a micturition diary for 7-days before the baseline and prior to each visit.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
micturitions
  Month 1: number analyzed (Participants) | 291 | 288 | 1158
  Month 1 | -1.09 (0.12) | -1.36 (0.12) | -1.64 (0.06)
  Month 3: number analyzed (Participants) | 282 | 288 | 1137
  Month 3 | -1.63 (0.13) | -1.87 (0.12) | 2.16 (0.06)
  Month 6: number analyzed (Participants) | 266 | 273 | 1107
  Month 6 | -1.85 (0.13) | -2.04 (0.13) | -2.39 (0.06)
  Month 9: number analyzed (Participants) | 264 | 261 | 1070
  Month 9 | -2.03 (0.13) | -2.03 (0.13) | -2.42 (0.06)
  Month 12: number analyzed (Participants) | 258 | 256 | 1048
  Month 12 | -2.20 (0.13) | -2.13 (0.14) | -2.64 (0.07)

16. Secondary Outcome: Number of Days With < 8 Micturitions Per Day During the 7-Day Micturition Diary Period Prior to Each Visit (at Months 1, 3, 6, 9, 12 and EoT)
Description: The number of days with < 8 micturitions was the number of valid diary days during the 7-day micturition diary period with with less than 8 micturitions per day.
Time Frame: Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point; LOCF was used for EoT.
Measure: Mean (Standard Error); unit: days
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
days
  Month 1: number analyzed (Participants) | 291 | 288 | 1158
  Month 1 | 1.90 (0.13) | 1.60 (0.12) | 2.08 (0.07)
  Month 3: number analyzed (Participants) | 282 | 288 | 1137
  Month 3 | 2.07 (0.14) | 2.14 (0.14) | 2.66 (0.08)
  Month 6: number analyzed (Participants) | 266 | 273 | 1107
  Month 6 | 2.35 (0.15) | 2.34 (0.15) | 2.87 (0.08)
  Month 9: number analyzed (Participants) | 264 | 261 | 1070
  Month 9 | 2.38 (0.16) | 2.33 (0.15) | 2.93 (0.08)
  Month 12: number analyzed (Participants) | 258 | 256 | 1048
  Month 12 | 2.61 (0.16) | 2.58 (0.16) | 3.17 (0.08)
  EoT: number analyzed (Participants) | 301 | 297 | 1184
  EoT | 2.52 (0.15) | 2.58 (0.15) | 3.10 (0.08)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio vs. Mirabegron 50 mg (EoT): Odds ratio was from a overdispersed binomial regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of micturitions per 24 hours as a covariate; Test type: Superiority; p = 0.002, Overdispersed Binomial Regression; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.14 to 1.8]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio vs. Solifenacin 5 mg (EoT): Odds ratio was from a overdispersed binomial regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of micturitions per 24 hours as a covariate; Test type: Superiority; p = 0.007, Overdispersed Binomial Regression; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.09 to 1.73]

17. Secondary Outcome: Change From Baseline to EoT in Corrected Micturition Frequency
Description: Corrected micturition frequency was defined as the mean number of micturitions per 24 hours that participants had at end of treatment if their fluid intake had remained unchanged since baseline. Corrected micturition frequency was calculated as the baseline mean volume voided per micturition multiplied by the baseline mean number of micturitions per 24 hours divided by the mean volume voided per micturition at EoT.
Time Frame: Baseline and Month 12
Population: FAS population; LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 301 | 297 | 1184
micturitions | -0.72 (0.17) | -1.11 (0.17) | -1.51 (0.08)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference vs. Mirabegron 50 mg (EoT): Difference of the adjusted mean was calculated by subtracting the adjusted mean of the mirabegron monotherapy group from the adjusted mean of the combination therapy group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as fixed factors and baseline mean number of micturitions per 24 hours as a covariate; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -0.78, 95% CI 2-sided [-1.16 to -0.41], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Difference vs. Solifenacin 5 mg (EoT): Difference of the adjusted mean was calculated by subtracting the adjusted mean of the solifenacin monotherapy group from the adjusted mean of the combination therapy group (solifenacin 5 mg + mirabegron 50 mg) based on the ANCOVA model with treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as fixed factors and baseline mean number of micturitions per 24 hours as a covariate; Test type: Superiority; p = 0.037, ANCOVA; Least Squares Mean Difference = -0.40, 95% CI 2-sided [-0.77 to -0.02], Standard Error of Mean 0.19

18. Secondary Outcome: Change From Baseline to Months 3, 6 and 12 in Mean Volume Voided Per Micturition
Description: The mean volume voided per micturition was calculated from the data recorded by the participant during 3 consecutive days with volume measurements during the 7-day micturition diary period prior to each visit.
Time Frame: Baseline and Months 3, 6, 12
Population: FAS population with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
mL
  Month 3: number analyzed (Participants) | 274 | 280 | 1125
  Month 3 | 15.34 (2.96) | 23.71 (2.92) | 34.89 (1.45)
  Month 6: number analyzed (Participants) | 265 | 268 | 1102
  Month 6 | 20.87 (3.21) | 27.08 (3.19) | 38.56 (1.57)
  Month 12: number analyzed (Participants) | 248 | 254 | 1028
  Month 12 | 21.85 (3.42) | 24.05 (3.37) | 38.72 (1.67)

19. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in Mean Number of Urgency Episodes (Grade 3 or 4) Per 24 Hours
Description: Urgency was defined as a complaint of a sudden, compelling desire to pass urine, which is difficult to defer. An urgency episode was defined as any micturition or incontinence episode recorded by the participant in the micturition diary for 7 days prior to each visit as 3 or 4 on the Patient Perception of Intensity of Urgency Scale (PPIUS), where 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could delay voiding a short while; 3 = Severe urgency, could not delay voiding; 4 = Urge incontinence, leaked before arriving to the toilet.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. Participants with ≥ 1 urgency episode at baseline were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
urgency episodes
  Month 1: number analyzed (Participants) | 291 | 288 | 1158
  Month 1 | -1.93 (0.17) | -2.31 (0.17) | -2.68 (0.09)
  Month 3: number analyzed (Participants) | 282 | 288 | 1137
  Month 3 | -2.68 (0.17) | -3.02 (0.17) | -3.36 (0.08)
  Month 6: number analyzed (Participants) | 266 | 273 | 1107
  Month 6 | -2.93 (0.17) | -3.17 (0.17) | -3.72 (0.08)
  Month 9: number analyzed (Participants) | 264 | 261 | 1070
  Month 9 | -3.40 (0.18) | -3.55 (0.18) | -3.87 (0.09)
  Month 12: number analyzed (Participants) | 258 | 256 | 1048
  Month 12 | -3.40 (0.17) | -3.56 (0.17) | -3.95 (0.09)
  EoT: number analyzed (Participants) | 301 | 297 | 1184
  EoT | -3.11 (0.17) | -3.45 (0.17) | -3.84 (0.08)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -0.73, 95% CI 2-sided [-1.10 to -0.37], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 12, analysis 2]; Test type: Superiority; p = 0.036, ANCOVA; Least Squares Mean Difference = -0.39, 95% CI 2-sided [-0.76 to -0.03], Standard Error of Mean 0.19

20. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in Mean Number of Nocturia Episodes Per 24 Hours
Description: A nocturia episode was defined as waking at night 1 or more times to void (i.e., any voiding associated with sleep disturbance between the time the participant goes to bed with the intention to sleep until the time the participant gets up in the morning with the intention to stay awake). The mean number of nocturia episodes was calculated from data recorded by the participant in the micturition diary for 7 days prior to each visit."
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. Only participants with ≥ 1 nocturia episode at baseline were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 262 | 252 | 1027
nocturia episodes
  Month 1: number analyzed (Participants) | 253 | 244 | 1000
  Month 1 | -0.20 (0.04) | -0.22 (0.04) | -0.34 (0.02)
  Month 3: number analyzed (Participants) | 247 | 244 | 985
  Month 3 | -0.34 (0.04) | -0.38 (0.04) | -0.46 (0.02)
  Month 6: number analyzed (Participants) | 231 | 231 | 958
  Month 6 | -0.41 (0.05) | -0.39 (0.05) | -0.49 (0.02)
  Month 9: number analyzed (Participants) | 229 | 221 | 927
  Month 9 | -0.42 (0.05) | -0.44 (0.05) | -0.50 (0.02)
  Month 12: number analyzed (Participants) | 225 | 217 | 906
  Month 12 | -0.46 (0.05) | -0.44 (0.05) | -0.56 (0.02)
  EoT: number analyzed (Participants) | 262 | 251 | 1023
  EoT | -0.45 (0.04) | -0.45 (0.04) | -0.55 (0.02)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.059, ANCOVA; Least Squares Mean Difference = -0.09, 95% CI 2-sided [-0.19 to 0.00], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 12, analysis 2]; Test type: Superiority; p = 0.068, ANCOVA; Least Squares Mean Difference = -0.09, 95% CI 2-sided [-0.19 to 0.01], Standard Error of Mean 0.05

21. Secondary Outcome: Number of Nocturia Episodes Reported During the 7-Day Micturition Diary Period Prior to Each Visit
Description: A nocturia episode was defined as waking at night 1 or more times to void (i.e., any voiding associated with sleep disturbance between the time the participant goes to bed with the intention to sleep until the time the participant gets up in the morning with the intention to stay awake). The number of nocturia episodes was the number of times a participant recorded a nocturia episode during the 7-day micturition diary period prior to each visit.
Time Frame: Months 1, 3, 6, 9, 12
Population: as for outcome 20
Measure: Mean (Standard Error); unit: nocturia episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 262 | 252 | 1027
nocturia episodes
  Month 1: number analyzed (Participants) | 253 | 244 | 1000
  Month 1 | 8.76 (0.41) | 9.23 (0.44) | 8.00 (0.20)
  Month 3: number analyzed (Participants) | 247 | 244 | 985
  Month 3 | 7.93 (0.39) | 7.92 (0.40) | 7.17 (0.19)
  Month 6: number analyzed (Participants) | 231 | 231 | 958
  Month 6 | 7.12 (0.35) | 7.86 (0.43) | 6.96 (0.20)
  Month 9: number analyzed (Participants) | 229 | 221 | 927
  Month 9 | 7.40 (0.38) | 7.48 (0.41) | 6.84 (0.20)
  Month 12: number analyzed (Participants) | 225 | 217 | 906
  Month 12 | 6.88 (0.38) | 7.39 (0.44) | 6.33 (0.19)
  EoT: number analyzed (Participants) | 262 | 251 | 1023
  EoT | 7.13 (0.37) | 7.47 (0.42) | 6.51 (0.19)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Rate ratio of number of nocturia episodes during the EoT 7-day diary between the combination therapy group and the mirabegron monotherapy group was calculated from a negative binomial regression model incl. treatment group, sex, age group (< 65, ≥ 65 years), geographic region and previous study history as factors, log(number of nocturia episodes divided by number of valid diary days) included as a covariate and post baseline number of valid diary days as the offset variable; Test type: Superiority; p = 0.067, Negative Binomial Regression; Rate Ratio = 0.90, 95% CI 2-sided [0.81 to 1.01], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Rate ratio of number of nocturia episodes during the EoT 7-day diary between the combination therapy group and the solifenacin monotherapy group was calculated from a negative binomial regression model incl. treatment group, sex, age group (< 65, ≥ 65 years), geographic region and previous study history as factors, log(number of nocturia episodes divided by number of valid diary days) included as a covariate and post baseline number of valid diary day as the offset variable; Test type: Superiority; p = 0.131, Negative Binomial Regression; Rate Ratio = 0.92, 95% CI [0.82 to 1.03], Standard Error of Mean 0.06

22. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in Number of Nocturia Episodes During the 7-Day Micturition Diary Period Prior to Each Visit
Description: as for outcome 21
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 262 | 252 | 1027
nocturia episodes
  Month 1: number analyzed (Participants) | 253 | 244 | 1000
  Month 1 | -1.56 (0.29) | -1.58 (0.29) | -2.39 (0.15)
  Month 3: number analyzed (Participants) | 247 | 244 | 985
  Month 3 | -2.45 (0.29) | -2.78 (0.30) | -3.26 (0.15)
  Month 6: number analyzed (Participants) | 231 | 231 | 958
  Month 6 | -3.08 (0.33) | -2.81 (0.33) | -3.44 (0.16)
  Month 9: number analyzed (Participants) | 229 | 221 | 927
  Month 9 | -2.91 (0.32) | -3.13 (0.32) | -3.55 (0.16)
  Month 12: number analyzed (Participants) | 225 | 217 | 906
  Month 12 | -3.29 (0.32) | -3.08 (0.33) | -3.97 (0.16)
  EoT: number analyzed (Participants) | 262 | 251 | 1023
  EoT | -3.24 (0.31) | -3.20 (0.32) | -3.90 (0.16)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.055, ANCOVA; Least Squares Mean Difference = -0.67, 95% CI 2-sided [-1.34 to 0.01], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 12, analysis 2]; Test type: Superiority; p = 0.048, ANCOVA; Least Squares Mean Difference = -0.70, 95% CI 2-sided [-1.39 to -0.01], Standard Error of Mean 0.35

23. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in Mean Number of Pads Used Per 24 Hours
Description: The mean number of pads used per 24 hours was calculated from data recorded by the participant in the micturition diary for 7 days prior to each visit.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. Only participants with ≥ 1 pads used at baseline were included in the analysis. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: pads
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 201 | 193 | 771
pads
  Month 1: number analyzed (Participants) | 193 | 185 | 741
  Month 1 | -0.67 (0.10) | -0.96 (0.11) | -1.25 (0.05)
  Month 3: number analyzed (Participants) | 188 | 184 | 734
  Month 3 | -1.12 (0.11) | -1.30 (0.11) | -1.49 (0.06)
  Month 6: number analyzed (Participants) | 174 | 173 | 712
  Month 6 | -1.30 (0.12) | -1.24 (0.12) | -1.59 (0.06)
  Month 9: number analyzed (Participants) | 173 | 166 | 689
  Month 9 | -1.38 (0.12) | -1.31 (0.13) | -1.65 (0.06)
  Month 12: number analyzed (Participants) | 170 | 162 | 678
  Month 12 | -1.35 (0.12) | -1.37 (0.13) | -1.67 (0.06)
  EoT: number analyzed (Participants) | 200 | 191 | 762
  EoT | -1.23 (0.12) | -1.38 (0.12) | -1.66 (0.06)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.002, ANCOVA; Least Squares Mean Difference = -0.42, 95% CI 2-sided [-0.69 to -0.16], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.039, ANCOVA; Least Squares Mean Difference = -0.28, 95% CI 2-sided [-0.55 to -0.01], Standard Error of Mean 0.14

24. Secondary Outcome: Number of Pads Used During the 7-Day Micturition Diary Period Prior to Each Visit
Description: The number of pads used was the number of times a participant recorded a new pad used during the 7-day micturition diary period prior to each visit.
Time Frame: Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. Only participants with ≥ 1 pad used at baseline were included in the analysis. LOCF was used for EoT.
Measure: Mean (Standard Error); unit: pads
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 201 | 193 | 771
pads
  Month 1: number analyzed (Participants) | 193 | 185 | 741
  Month 1 | 12.67 (1.98) | 12.55 (1.59) | 8.75 (0.50)
  Month 3: number analyzed (Participants) | 188 | 184 | 734
  Month 3 | 9.61 (1.12) | 9.47 (1.28) | 7.23 (0.5)
  Month 6: number analyzed (Participants) | 174 | 173 | 712
  Month 6 | 7.99 (1.03) | 9.16 (1.28) | 6.51 (0.47)
  Month 9: number analyzed (Participants) | 173 | 166 | 689
  Month 9 | 7.65 (1.08) | 8.91 (1.28) | 6.18 (0.46)
  Month 12: number analyzed (Participants) | 170 | 162 | 678
  Month 12 | 7.60 (1.05) | 8.09 (1.23) | 5.70 (0.44)
  EoT: number analyzed (Participants) | 200 | 191 | 762
  EoT | 9.09 (1.07) | 8.54 (1.10) | 6.33 (0.45)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Rate ratio vs. Mirabegron 50 mg (EoT): Rate ratio of number of pads during the EoT 7-day diary between the combination therapy group and the mirabegron monotherapy group is calculated from a negative binomial regression model incl. treatment group, sex, age group (< 65, ≥ 65 years), geographic region and previous study history as factors, log(number of pads divided by number of valid diary days) included as a covariate and post baseline number of valid diary days as the offset variable; Test type: Superiority; p < 0.001, Negative Binomial Regression; Rate Ratio = 0.58, 95% CI 2-sided [0.45 to 0.76], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Rate ratio vs. Solifenacin 5 mg (EoT): Rate ratio of number of pads during the EoT 7-day diary between the combination therapy group and the solifenacin monotherapy group is calculated from a negative binomial regression model incl. treatment group, sex, age group (< 65, ≥ 65 years), geographic region and previous study history as factors, log(number of pads divided by number of valid diary days) included as a covariate and post baseline number of valid diary days as the offset variable; Test type: Superiority; p = 0.044, Negative Binomial Regression; Rate Ratio = 0.76, 95% CI 2-sided [0.58 to 0.99], Standard Error of Mean 0.14

25. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in Number of Pads Used During the 7-Day Micturition Diary Period Prior to Each Visit
Description: as for outcome 24
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: pads
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 201 | 193 | 771
pads
  Month 1: number analyzed (Participants) | 193 | 185 | 741
  Month 1 | -4.74 (0.71) | -6.72 (0.72) | -8.89 (0.36)
  Month 3: number analyzed (Participants) | 188 | 184 | 734
  Month 3 | -7.83 (0.77) | -9.21 (0.78) | 10.47 (0.39)
  Month 6: number analyzed (Participants) | 174 | 173 | 712
  Month 6 | -9.09 (0.85) | -8.86 (0.85) | -11.12 (0.42)
  Month 9: number analyzed (Participants) | 173 | 166 | 689
  Month 9 | -9.59 (0.87) | -9.33 (0.89) | -11.44 (0.43)
  Month 12: number analyzed (Participants) | 170 | 162 | 678
  Month 12 | -9.39 (0.85) | -9.92 (0.87) | -11.66 (0.42)
  EoT: number analyzed (Participants) | 200 | 191 | 762
  EoT | -8.59 (0.82) | -9.89 (0.84) | -11.58 (0.42)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.001, ANCOVA; Least Squares Mean Difference = -2.98, 95% CI 2-sided [-4.78 to -1.18], Standard Error of Mean 0.92
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.072, ANCOVA; Least Squares Mean Difference = -1.68, 95% CI 2-sided [-3.52 to 0.15], Standard Error of Mean 0.93

26. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9 and 12 in the OAB-q Symptom Bother Score
Description: as for outcome 5
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
units on a scale
  Month 1: number analyzed (Participants) | 281 | 286 | 1132
  Month 1 | -16.37 (1.08) | -20.82 (1.07) | -22.86 (0.54)
  Month 3: number analyzed (Participants) | 278 | 286 | 1137
  Month 3 | -19.69 (1.08) | -23.13 (1.07) | -26.88 (0.53)
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | -20.97 (1.14) | -24.27 (1.12) | -27.73 (0.55)
  Month 9: number analyzed (Participants) | 261 | 264 | 1077
  Month 9 | -21.41 (1.15) | -25.82 (1.14) | -28.45 (0.56)
  Month 12: number analyzed (Participants) | 250 | 255 | 1049
  Month 12 | -23.41 (1.19) | -25.38 (1.18) | -30.18 (0.58)

27. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in Health-Related Quality of Life Questionnaire (HRQoL): Total Score
Description: The OAB-q is a self-reported questionnaire with items relating to symptom bother and HRQoL. The HRQoL portion consists of 25 HRQoL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each item was scored 1-6. The total score was calculated by adding the 4 HRQoL subscale scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
units on a scale
  Month 1: number analyzed (Participants) | 281 | 286 | 1132
  Month 1 | 11.67 (0.92) | 14.01 (0.91) | 15.69 (0.45)
  Month 3: number analyzed (Participants) | 278 | 286 | 1137
  Month 3 | 15.25 (0.95) | 16.41 (0.94) | 19.26 (0.47)
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | 16.63 (1.02) | 17.96 (1.00) | 20.03 (0.49)
  Month 9: number analyzed (Participants) | 261 | 264 | 1077
  Month 9 | 16.69 (1.02) | 18.53 (1.01) | 20.75 (0.50)
  Month 12: number analyzed (Participants) | 250 | 255 | 1049
  Month 12 | 17.33 (1.04) | 18.80 (1.03) | 21.82 (0.51)
  EoT: number analyzed (Participants) | 290 | 294 | 1163
  EoT | 16.57 (1.00) | 18.47 (0.99) | 21.33 (0.50)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = 4.76, 95% CI 2-sided [2.56 to 6.96], Standard Error of Mean 1.12
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.010, ANCOVA; Least Squares Mean Difference = 2.86, 95% CI 2-sided [0.68 to 5.04], Standard Error of Mean 1.11

28. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in HRQoL Subscale Score: Coping
Description: The OAB-q is a self-reported questionnaire with items relating to symptom bother and HRQoL. The HRQoL portion consists of 25 HRQoL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each item was scored 1-6. HRQoL subscales (coping, concern, sleep and social) and total score were transformed to range from 0 (worst quality of life) to 100 (best quality of life), with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
units on a scale
  Month 1: number analyzed (Participants) | 281 | 286 | 1132
  Month 1 | 13.05 (1.09) | 15.40 (1.08) | 17.58 (0.54)
  Month 3: number analyzed (Participants) | 278 | 286 | 1137
  Month 3 | 17.57 (1.14) | 18.38 (1.13) | 21.64 (0.56)
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | 19.68 (1.22) | 20.53 (1.19) | 22.73 (0.59)
  Month 9: number analyzed (Participants) | 261 | 264 | 1077
  Month 9 | 19.54 (1.21) | 21.21 (1.20) | 23.58 (0.59)
  Month 12: number analyzed (Participants) | 250 | 255 | 1049
  Month 12 | 19.47 (1.25) | 21.90 (1.23) | 24.86 (0.61)
  EoT: number analyzed (Participants) | 290 | 294 | 1163
  EoT | 18.54 (1.19) | 21.13 (1.18) | 24.14 (0.59)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = 5.60, 95% CI 2-sided [2.99 to 8.20], Standard Error of Mean 1.33
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.022, ANCOVA; Least Squares Mean Difference = 3.01, 95% CI 2-sided [0.43 to 5.60], Standard Error of Mean 1.32

29. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in HRQoL Subscale Score: Concern
Description: as for outcome 28
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
units on a scale
  Month 1: number analyzed (Participants) | 281 | 286 | 1132
  Month 1 | 13.24 (1.03) | 15.49 (1.02) | 17.60 (0.51)
  Month 3: number analyzed (Participants) | 278 | 286 | 1137
  Month 3 | 16.37 (1.05) | 17.64 (1.04) | 21.23 (0.52)
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | 17.77 (1.10) | 19.05 (1.07) | 21.73 (0.53)
  Month 9: number analyzed (Participants) | 261 | 264 | 1077
  Month 9 | 18.15 (1.11) | 19.74 (1.10) | 22.30 (0.54)
  Month 12: number analyzed (Participants) | 250 | 255 | 1049
  Month 12 | 19.10 (1.12) | 19.40 (1.10) | 23.30 (0.54)
  EoT: number analyzed (Participants) | 290 | 294 | 1163
  EoT | 17.98 (1.08) | 19.22 (1.07) | 23.00 (0.54)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = 5.01, 95% CI 2-sided [2.65 to 7.38], Standard Error of Mean 1.21
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.002, ANCOVA; Least Squares Mean Difference = 3.78, 95% CI 2-sided [1.43 to 6.13], Standard Error of Mean 1.20

30. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in HRQoL Subscale Score: Sleep
Description: The OAB-q is a self-reported questionnaire with items relating to symptom bother and HRQoL. The HRQoL portion consisted of 25 HRQoL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each time was scored 1-6. HRQoL subscales (coping, concern, sleep and social) and total score were transformed to range from 0 (worst quality of life) to 100 (best quality of life), with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
units on a scale
  Month 1: number analyzed (Participants) | 281 | 286 | 1132
  Month 1 | 10.96 (1.08) | 14.24 (1.07) | 15.82 (0.54)
  Month 3: number analyzed (Participants) | 278 | 286 | 1137
  Month 3 | 14.09 (1.12) | 16.71 (1.10) | 19.75 (0.55)
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | 14.84 (1.22) | 17.70 (1.19) | 20.09 (0.59)
  Month 9: number analyzed (Participants) | 261 | 264 | 1077
  Month 9 | 14.86 (1.22) | 17.73 (1.21) | 21.15 (0.60)
  Month 12: number analyzed (Participants) | 250 | 255 | 1049
  Month 12 | 16.53 (1.29) | 18.28 (1.27) | 22.17 (0.63)
  EoT: number analyzed (Participants) | 290 | 294 | 1163
  EoT | 16.44 (1.22) | 18.32 (1.21) | 21.59 (0.61)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = 5.15, 95% CI 2-sided [2.47 to 7.83], Standard Error of Mean 1.36
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.016, ANCOVA; Least Squares Mean Difference = 3.27, 95% CI 2-sided [0.62 to 5.93], Standard Error of Mean 1.35

31. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in HRQL Subscale Score: Social
Description: as for outcome 28
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
units on a scale
  Month 1: number analyzed (Participants) | 281 | 286 | 1132
  Month 1 | 7.99 (0.84) | 9.41 (0.83) | 9.89 (0.42)
  Month 3: number analyzed (Participants) | 278 | 286 | 1137
  Month 3 | 11.14 (0.85) | 11.19 (0.84) | 12.22 (0.42)
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | 11.89 (0.89) | 12.54 (0.87) | 13.30 (0.43)
  Month 9: number analyzed (Participants) | 261 | 264 | 1077
  Month 9 | 11.92 (0.90) | 13.33 (0.89) | 13.64 (0.44)
  Month 12: number analyzed (Participants) | 250 | 255 | 1049
  Month 12 | 12.25 (0.90) | 13.47 (0.89) | 14.52 (0.44)
  EoT: number analyzed (Participants) | 290 | 294 | 1163
  EoT | 11.57 (0.87) | 13.22 (0.87) | 14.25 (0.43)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.006, ANCOVA; Least Squares Mean Difference = 2.68, 95% CI 2-sided [0.77 to 4.59], Standard Error of Mean 0.98
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.287, ANCOVA; Least Squares Mean Difference = 1.03, 95% CI 2-sided [-0.87 to 2.93], Standard Error of Mean 0.97

32. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9 and 12 in the Patient's Assessment of TS-VAS
Description: as for outcome 6
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
units on a scale
  Month 1: number analyzed (Participants) | 280 | 286 | 1131
  Month 1 | 1.88 (0.12) | 1.95 (0.12) | 2.27 (0.06)
  Month 3: number analyzed (Participants) | 277 | 286 | 1136
  Month 3 | 2.10 (0.11) | 2.06 (0.11) | 2.57 (0.06)
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | 2.22 (0.12) | 2.25 (0.12) | 2.72 (0.06)
  Month 9: number analyzed (Participants) | 261 | 263 | 1076
  Month 9 | 2.24 (0.12) | 2.28 (0.12) | 2.74 (0.06)
  Month 12: number analyzed (Participants) | 250 | 255 | 1049
  Month 12 | 2.33 (0.12) | 2.34 (0.12) | 2.89 (0.06)

33. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in Patient Perception of Bladder Condition (PPBC)
Description: The PPBC is a validated, global assessment tool using a 6-point Likert scale on which participants rated their subjective impression of their current bladder condition. Participants assessed their bladder condition using this scale: 1. Does not cause me any problems at all; 2. Causes me some very minor problems; 3. Causes me some minor problems; 4. Causes me (some) moderate problems; 5. Causes me severe problems; 6. Causes me many severe problems.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
units on a scale
  Month 1: number analyzed (Participants) | 281 | 287 | 1133
  Month 1 | -0.84 (0.07) | -0.89 (0.07) | -1.05 (0.03)
  Month 3: number analyzed (Participants) | 278 | 286 | 1137
  Month 3 | -1.09 (0.07) | -1.08 (0.07) | -1.33 (0.03)
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | -1.11 (0.07) | -1.18 (0.07) | -1.42 (0.04)
  Month 9: number analyzed (Participants) | 261 | 264 | 1077
  Month 9 | -1.25 (0.07) | -1.31 (0.07) | -1.48 (0.04)
  Month 12: number analyzed (Participants) | 251 | 255 | 1049
  Month 12 | -1.29 (0.08) | -1.36 (0.07) | -1.59 (0.04)
  EoT: number analyzed (Participants) | 290 | 294 | 1163
  EoT | -1.22 (0.07) | -1.34 (0.07) | -1.54 (0.04)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -0.32, 95% CI 2-sided [-0.47 to -0.16], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.011, ANCOVA; Least Squares Mean Difference = -0.20, 95% CI 2-sided [-0.36 to -0.05], Standard Error of Mean 0.08

34. Secondary Outcome: Percentage of Participants in Each Category of Patient's Global Impression of Change (PGIC) Scale: Impression in Bladder Symptoms at Month 12 and EoT
Description: The PGIC is a 2-part questionnaire, assessing both the change in the patient's overall condition and change in bladder condition since the start of the study (from very much worse to very much improved).
Time Frame: Month 12
Population: FAS population with data available. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 12: Very much improved | 25.5 | 23.4 | 33.8
  Month 12: Much improved | 30.5 | 35.8 | 34.0
  Month 12: Minimally improved | 21.9 | 19.7 | 16.1
  Month 12: No change | 5.0 | 6.4 | 4.5
  Month 12: Minimally worse | 0.7 | 0.7 | 0.4
  Month 12: Much worse | 1.0 | 0.3 | 0.1
  Month 12: Very much worse | 0.3 | 0.3 | 0.5
  EoT: Very much improved | 25.8 | 24.4 | 34.1
  EoT: Much improved | 31.5 | 37.1 | 34.7
  EoT: Minimally improved | 22.2 | 20.4 | 16.6
  EoT: No change | 6.3 | 7.0 | 5.1
  EoT: Minimally worse | 0.7 | 0.7 | 0.4
  EoT: Much worse | 1.3 | 0.7 | 0.1
  EoT: Very much worse | 0.3 | 0.3 | 0.5

35. Secondary Outcome: Percentage of Participants in Each Category of PGIC Scale: Impression in General Health at Month 12 and EoT
Description: as for outcome 34
Time Frame: Month 12
Population: FAS population with data available. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 12: Very much improved | 12.9 | 14.7 | 18.0
  Month 12: Much improved | 23.8 | 26.8 | 28.7
  Month 12: Minimally improved | 18.9 | 17.1 | 18.7
  Month 12: No change | 24.2 | 24.7 | 20.7
  Month 12: Minimally worse | 3.6 | 2.7 | 2.7
  Month 12: Much worse | 0.7 | 0 | 0.4
  Month 12: Very much worse | 0.7 | 0.7 | 0.3
  EoT: Very much improved | 13.2 | 15.1 | 18.3
  EoT: Much improved | 24.5 | 27.8 | 28.9
  EoT: Minimally improved | 19.2 | 18.1 | 19.1
  EoT: No change | 25.8 | 25.8 | 21.6
  EoT: Minimally worse | 3.6 | 3.0 | 2.8
  EoT: Much worse | 1.0 | 0.3 | 0.5
  EoT: Very much worse | 0.7 | 0.7 | 0.3

36. Secondary Outcome: Number of Participants With Change From Baseline to EoT in European Quality of Llife in 5 Dimensions (EQ-5D) Questionnaire Subscale Score: Mobility
Description: The EQ-5D questionnaire is an international, standardized, nondisease specific instrument for describing and valuing health status, and has 5 dimensions: Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has 5 response levels ranging from level 1 (no problem or none) to level 5 (unable to perform activity).
Time Frame: Baseline and 12 Months
Population: FAS population; LOCF was used for EoT.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
Participants
  No problems -> no problems | 164 | 164 | 675
  No problems -> slight problems | 15 | 15 | 56
  No problems -> moderate problems | 10 | 4 | 26
  No problems -> severe problems | 1 | 1 | 2
  No problems -> unable to walk about | 1 | 0 | 0
  No problems -> no data | 3 | 0 | 7
  Slight problems -> no problems | 19 | 24 | 83
  Slight problems -> slight problems | 18 | 29 | 87
  Slight problems -> moderate problems | 4 | 6 | 26
  Slight problems -> severe problems | 3 | 1 | 2
  Slight problems -> unable to walk about | 0 | 0 | 0
  Slight problems -> no data | 2 | 1 | 0
  Moderate problems -> no problems | 14 | 11 | 38
  Moderate problems -> slight problems | 13 | 17 | 47
  Moderate problems -> moderate problems | 9 | 5 | 50
  Moderate problems -> severe problems | 2 | 4 | 8
  Moderate problems -> unable to walk about | 0 | 0 | 0
  Moderate problems -> no data | 0 | 0 | 1
  Severe problems -> no problems | 2 | 4 | 15
  Severe problems -> slight problems | 2 | 2 | 13
  Severe problems -> moderate problems | 6 | 4 | 16
  Severe problems -> severe problems | 5 | 3 | 15
  Severe problems -> unable to walk about | 1 | 0 | 2
  Severe problems -> no data | 0 | 0 | 0
  Unable to walk about -> no problems | 0 | 0 | 1
  Unable to walk about -> slight problems | 0 | 0 | 1
  Unable to walk about -> moderate problems | 0 | 0 | 0
  Unable to walk about -> severe problems | 0 | 0 | 0
  Unable to walk about -> unable to walk about | 0 | 0 | 0
  Unable to walk about -> no data | 0 | 0 | 0
  No data -> no problems | 4 | 3 | 19
  No data -> slight problems | 4 | 1 | 3
  No data -> moderate problems | 0 | 0 | 0
  No data -> severe problems | 0 | 0 | 0
  No data -> unable to walk about | 0 | 0 | 0
  No data -> no data | 0 | 0 | 0

37. Secondary Outcome: Number of Participants With Change From Baseline to EoT in EQ-5D Questionnaire Subscale Score: Self-care
Description: as for outcome 36
Time Frame: Baseline and Month 12
Population: FAS populaton; LOCF was used for EoT.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
Participants
  No problems -> no problems | 223 | 232 | 906
  No problems -> slight problems | 12 | 9 | 40
  No problems -> moderate problems | 8 | 0 | 12
  No problems -> severe problems | 0 | 1 | 2
  No problems -> unable to wash/dress myself | 0 | 0 | 0
  No problems -> no data | 5 | 1 | 7
  Slight problems -> no problems | 16 | 18 | 64
  Slight problems -> slight problems | 9 | 14 | 44
  Slight problems -> moderate problems | 0 | 4 | 12
  Slight problems -> severe problems | 0 | 1 | 1
  Slight problems -> unable to wash/dress myself | 0 | 0 | 0
  Slight problems -> no data | 0 | 0 | 1
  Moderate problems -> no problems | 5 | 4 | 18
  Moderate problems -> slight problems | 5 | 6 | 20
  Moderate problems -> moderate problems | 5 | 3 | 21
  Moderate problems -> severe problems | 0 | 0 | 2
  Moderate problems -> unable to wash/dress myself | 0 | 0 | 0
  Moderate problems -> no data | 0 | 0 | 0
  Severe problems -> no problems | 0 | 1 | 8
  Severe problems -> slight problems | 1 | 0 | 3
  Severe problems -> moderate problems | 3 | 1 | 4
  Severe problems -> severe problems | 1 | 0 | 5
  Severe problems -> unable to wash/dress myself | 0 | 0 | 0
  Severe problems -> no data | 0 | 0 | 0
  Unable to wash/dress myself -> no problems | 0 | 0 | 0
  Unable to wash/dress myself -> slight problems | 0 | 0 | 1
  Unable to wash/dress myself -> moderate problems | 0 | 0 | 0
  Unable to wash/dress myself -> severe problems | 0 | 0 | 0
  Unable to wash/dress myself -> unable to wash/dres | 1 | 0 | 0
  Unable to wash/dress myself -> no data | 0 | 0 | 0
  No data -> no problems | 6 | 3 | 22
  No data -> slight problems | 2 | 1 | 0
  No data -> moderate problems | 0 | 0 | 0
  No data -> severe problems | 0 | 0 | 0
  No data -> unable to wash/dress myself | 0 | 0 | 0
  No data -> no data | 0 | 0 | 0

38. Secondary Outcome: Number of Participants With Change From Baseline to EoT in EQ-5D Questionnaire Subscale Score: Usual Activities
Description: as for outcome 36
Time Frame: Baseline and Month 12
Population: FAS population; LOCF was used for EoT.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
Participants
  No problems -> No problems | 165 | 160 | 672
  No problems -> Slight problems | 13 | 16 | 65
  No problems -> Moderate problems | 8 | 4 | 15
  No problems -> Severe problems | 1 | 0 | 1
  No problems -> unable to do usual activities | 0 | 0 | 0
  No problems -> no data | 4 | 0 | 7
  Slight problems -> no problems | 27 | 39 | 131
  Slight problems -> slight problems | 28 | 33 | 85
  Slight problems -> moderate problems | 5 | 6 | 26
  Slight problems -> severe problems | 2 | 1 | 1
  Slight problems ->unable to do usual activities | 0 | 0 | 0
  Slight problems -> no data | 1 | 0 | 0
  Moderate problems -> no problems | 12 | 12 | 40
  Moderate problems -> slight problems | 11 | 9 | 44
  Moderate problems -> moderate problems | 7 | 4 | 43
  Moderate problems -> severe problems | 2 | 0 | 2
  Moderate problems ->unable to do usual activities | 0 | 0 | 0
  Moderate problems -> no data | 0 | 1 | 1
  Severe problems -> no problems | 2 | 1 | 10
  Severe problems -> slight problems | 0 | 2 | 9
  Severe problems -> moderate problems | 0 | 6 | 7
  Severe problems -> severe problems | 4 | 1 | 6
  Severe problems -> unable to do usual activities | 0 | 0 | 1
  Severe problems -> no data | 0 | 0 | 0
  Unable to do usual activities -> no problems | 0 | 0 | 0
  Unable to do usual activities -> slight problems | 0 | 0 | 1
  Unable to do usual activities -> moderate problems | 1 | 0 | 4
  Unable to do usual activities -> severe problems | 0 | 0 | 0
  Unable to do usual activities -> unable to do | 1 | 0 | 0
  Unable to do usual activities -> no data | 0 | 0 | 0
  No data -> no problems | 6 | 2 | 20
  No data -> slight problems | 1 | 2 | 2
  No data -> moderate problems | 1 | 0 | 0
  No data -> severe problems | 0 | 0 | 0
  No data -> unable to do usual activities | 0 | 0 | 0
  No data -> no data | 0 | 0 | 0

39. Secondary Outcome: Number of Participants With Change From Baseline to EoT in EQ-5D Questionnaire Subscale Score: Pain/Discomfort
Description: The EQ-5D questionnaire is an international, standardized, nondisease specific instrument for describing and valuing health status, and had 5 dimensions: Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has 5 response levels ranging from level 1 (no problem or none) to level 5 (unable to perform activity).
Time Frame: Baseline and Month 12
Population: FAS population; LOCF was used for EoT.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
Participants
  No pain/discomfort -> no pain/discomfort | 120 | 119 | 495
  No pain/discomfort -> slight pain/discomfort | 21 | 19 | 70
  No pain/discomfort -> moderate pain/discomfort | 7 | 1 | 20
  No pain/discomfort -> severe pain/discomfort | 1 | 0 | 3
  No pain/discomfort -> extreme pain/discomfort | 0 | 0 | 0
  No pain/discomfort -> no data | 2 | 1 | 6
  Slight pain/discomfort -> no pain/discomfort | 44 | 37 | 132
  Slight pain/discomfort -> slight pain/discomfort | 24 | 48 | 152
  Slight pain/discomfort -> moderate pain/discomfort | 11 | 9 | 26
  Slight pain/discomfort -> severe pain/discomfort | 2 | 1 | 5
  Slight pain/discomfort -> extreme pain/discomfort | 0 | 0 | 1
  Slight pain/discomfort -> no data | 0 | 0 | 1
  Moderate pain/discomfort -> no pain/discomfort | 9 | 11 | 49
  Moderate pain/discomfort -> slight pain/discomfort | 19 | 17 | 78
  Moderate pain/discomfort -> moderate pain/discomf | 16 | 10 | 65
  Moderate pain/discomfort -> severe pain/discomfort | 2 | 3 | 8
  Moderate pain/discomfort -> extreme pain/discomf | 0 | 0 | 1
  Moderate pain/discomfort -> no data | 1 | 0 | 1
  Severe pain/discomfort -> no pain/discomfort | 3 | 6 | 15
  Severe pain/discomfort -> slight pain/discomfort | 2 | 3 | 9
  Severe pain/discomfort -> moderate pain/discomfort | 5 | 5 | 13
  Severe pain/discomfort -> severe pain/discomfort | 2 | 3 | 11
  Severe pain/discomfort -> extreme pain/discomfort | 0 | 0 | 1
  Severe pain/discomfort -> no data | 1 | 0 | 0
  Extreme pain/discomfort -> no pain/discomfort | 0 | 0 | 0
  Extreme pain/discomfort -> slight pain/discomfort | 0 | 0 | 3
  Extreme pain/discomfort -> moderate pain/discomf | 1 | 0 | 2
  Extreme pain/discomfort -> severe pain/discomfort | 0 | 2 | 2
  Extreme pain/discomfort -> extreme pain/discomfort | 0 | 0 | 2
  Extreme pain/discomfort -> no data | 1 | 0 | 0
  No data -> no pain/discomfort | 5 | 1 | 11
  No data -> slight pain/discomfort | 3 | 3 | 11
  No data -> moderate pain/discomfort | 0 | 0 | 0
  No data -> extreme pain/discomfort | 0 | 0 | 0
  No data -> severe pain/discomfort | 0 | 0 | 0
  No data -> no data | 0 | 0 | 0

40. Secondary Outcome: Number of Participants With Change From Baseline to EoT in EQ-5D Questionnaire Subscale Score: Anxiety/Depression
Description: as for outcome 39
Time Frame: Baseline and Month 12
Population: FAS population; LOCF was used for EoT.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
Participants
  Not anxious -> not anxious | 137 | 142 | 588
  Not anxious -> slightly anxious | 22 | 18 | 68
  Not anxious -> moderately anxious | 4 | 1 | 7
  Not anxious -> severely anxious | 1 | 0 | 1
  Not anxious -> extremely anxious | 0 | 0 | 0
  Not anxious -> no data | 3 | 1 | 5
  Slightly anxious -> not anxious | 35 | 43 | 177
  Slightly anxious -> slightly anxious | 30 | 33 | 106
  Slightly anxious -> moderately anxious | 4 | 8 | 21
  Slightly anxious -> severely anxious | 3 | 1 | 0
  Slightly anxious -> extremely anxious | 0 | 1 | 1
  Slightly anxious -> no data | 1 | 0 | 1
  Moderately anxious -> not anxious | 15 | 11 | 37
  Moderately anxious -> slightly anxious | 11 | 14 | 55
  Moderately anxious -> moderately anxious | 12 | 8 | 35
  Moderately anxious -> severely anxious | 1 | 1 | 5
  Moderately anxious -> extremely anxious | 0 | 0 | 0
  Moderately anxious -> no data | 0 | 0 | 1
  Severely anxious -> not anxious | 2 | 2 | 10
  Severely anxious -> slightly anxious | 3 | 2 | 14
  Severely anxious -> moderately anxious | 5 | 3 | 13
  Severely anxious -> severely anxious | 2 | 1 | 7
  Severely anxious -> extremely anxious | 1 | 0 | 1
  Severely anxious -> no data | 1 | 0 | 1
  Extremely anxious -> not anxious | 0 | 1 | 4
  Extremely anxious -> slightly anxious | 0 | 2 | 2
  Extremely anxious -> moderately anxious | 1 | 0 | 8
  Extremely anxious -> severely anxious | 0 | 2 | 2
  Extremely anxious -> extremely anxious | 0 | 0 | 1
  Extremely anxious -> no data | 0 | 0 | 0
  No data -> not anxious | 6 | 3 | 14
  No data -> slightly anxious | 1 | 1 | 7
  No data -> moderately anxious | 1 | 0 | 0
  No data -> severely anxious | 0 | 0 | 0
  No data -> extremely anxious | 0 | 0 | 1
  No data -> no data | 0 | 0 | 0

41. Secondary Outcome: Change From Baseline to Months 6, 12 and EoT in Work Productivity and Activity Impairment: Specific Health Problem Questionnaire (WPAI:SHP) Score: Percent Work Time Missed
Description: The WPAI:SHP is a self-administered questionnaire with 6 questions (Q1=Employment status; Q2=Hours absent from work due to the bladder condition; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the bladder condition on productivity while working; Q6=Impact of the bladder condition on productivity while doing regular daily activities other than work) and a 1-week recall period. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. A negative change from baseline indicated improvement.
Time Frame: Baseline and Months 6,12
Population: FAS population with data available at each time point. Only participants with both baseline and post-baseline values and who were employed during the study are included in the analysis. LOCF was used for EoT.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 114 | 136 | 468
percentage of work time missed
  Month 6: number analyzed (Participants) | 86 | 112 | 379
  Month 6 | -0.49 (17.12) | -0.59 (15.67) | -3.11 (20.68)
  Month 12: number analyzed (Participants) | 83 | 110 | 359
  Month 12 | 0.39 (15.55) | -1.95 (18.51) | -3.74 (23.83)
  EoT: number analyzed (Participants) | 96 | 124 | 421
  EoT | -0.45 (18.51) | -1.30 (18.04) | -3.26 (22.88)

42. Secondary Outcome: Change From Baseline to Months 6, 12 and EoT in WPAI:SHP Score: Percent Impairment While Working
Description: as for outcome 41
Time Frame: Baseline and Months 6, 12
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 114 | 135 | 461
percentage of impairment while working
  Month 6: number analyzed (Participants) | 85 | 111 | 372
  Month 6 | -16.94 (24.10) | -12.97 (21.05) | -13.41 (24.37)
  Month 12: number analyzed (Participants) | 83 | 108 | 349
  Month 12 | -19.16 (23.38) | -14.72 (27.32) | -16.68 (24.16)
  EoT: number analyzed (Participants) | 96 | 123 | 414
  EoT | -17.81 (23.45) | -13.90 (27.18) | -15.63 (25.61)

43. Secondary Outcome: Change From Baseline to Months 6, 12 in WPAI:SHP Score: Percent Overall Work Impairment
Description: The WPAI:SHP is a self-administered questionnaire with 6 questions (Q1=Employment status; Q2=Hours absent from work due to the bladder condition; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the bladder condition on productivity while working; Q6=Impact of the bladder condition on productivity while doing regular daily activities other than work) and a 1-week recall period. WPAI outcomes arre expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. A negative change from baseline indicated improvement.
Time Frame: Baseline and Months 6, 12
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: percentage of overall work impairment
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 114 | 135 | 461
percentage of overall work impairment
  Month 6: number analyzed (Participants) | 85 | 111 | 372
  Month 6 | -16.33 (27.58) | -12.09 (22.26) | -13.99 (26.04)
  Month 12: number analyzed (Participants) | 83 | 108 | 349
  Month 12 | -17.83 (26.90) | -15.38 (27.97) | -17.27 (27.25)
  EoT: number analyzed (Participants) | 96 | 123 | 414
  EoT | -16.83 (27.63) | -14.16 (27.51) | -16.15 (28.51)

44. Secondary Outcome: Change From Baseline to Months 6, 12 in WPAI:SHP Score: Percent Activity Impairment
Description: as for outcome 41
Time Frame: Baseline and Months 6, 12
Population: FAS population with data available at each time point. Only participants with both baseline and post-baseline values during the study are included in the analysis. LOCF was used for EoT.
Measure: Mean (Standard Deviation); unit: percentage of activity Impairment
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 292 | 285 | 1167
percentage of activity Impairment
  Month 6: number analyzed (Participants) | 258 | 272 | 1105
  Month 6 | -15.04 (27.08) | -16.25 (24.78) | -16.94 (28.49)
  Month 12: number analyzed (Participants) | 248 | 255 | 1045
  Month 12 | -16.85 (27.57) | -14.12 (29.87) | -18.91 (29.26)
  EoT: number analyzed (Participants) | 274 | 281 | 1124
  EoT | -16.02 (27.63) | -14.02 (30.29) | -18.75 (29.14)

45. Secondary Outcome: Percentage of Participants With Zero Incontinence Episodes Per 24 Hours Using the Last 3 Diary Days at Months 1, 3, 6, 9, 12 and EoT
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The percentage of participants with no incontinence episodes recorded during the last 3 days of the 7-day micturition diary is reported.
Time Frame: Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 291 | 288 | 1158
  Month 1 | 24.4 | 39.9 | 38.3
  Month 3: number analyzed (Participants) | 282 | 288 | 1137
  Month 3 | 40.1 | 44.8 | 49.6
  Month 6: number analyzed (Participants) | 266 | 273 | 1107
  Month 6 | 40.6 | 50.5 | 54.7
  Month 9: number analyzed (Participants) | 264 | 261 | 1070
  Month 9 | 47.0 | 54.4 | 55.8
  Month 12: number analyzed (Participants) | 258 | 256 | 1048
  Month 12 | 51.6 | 55.5 | 61.2
  EoT: number analyzed (Participants) | 301 | 297 | 1184
  EoT | 47.8 | 53.2 | 58.8
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio was from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of incontinence episodes per 24 hours during the last 3 days as a covariate; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.26 to 2.15]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 45, analysis 1]; Test type: Superiority; p = 0.080, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.97 to 1.67]

46. Secondary Outcome: Percentage of Participants With ≥ 10 Points Improvement From Baseline in the OAB-q Symptom Bother Score at Months 1, 3, 6, 9, 12 and EoT
Description: The OAB-q is a self-reported questionnaire with items relating to symptom bother and HRQoL. The symptom bother portion consists of 8 items, rated on a 6-point Likert scale (1 through 6). The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 (least severity) to 100 (worst severity). A negative change from baseline indicated an improvement.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 281 | 286 | 1132
  Month 1 | 63.7 | 67.5 | 72.8
  Month 3: number analyzed (Participants) | 278 | 286 | 1137
  Month 3 | 69.1 | 71.3 | 81.8
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | 70.4 | 74.6 | 80.5
  Month 9: number analyzed (Participants) | 261 | 264 | 1077
  Month 9 | 70.1 | 76.1 | 82.9
  Month 12: number analyzed (Participants) | 250 | 255 | 1049
  Month 12 | 72.8 | 74.1 | 84.4
  EoT: number analyzed (Participants) | 290 | 294 | 1163
  EoT | 70.7 | 72.4 | 82.9
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio was from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline OAB-q subscale as a covariate; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.49 to 2.78]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 46, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.37 to 2.57]

47. Secondary Outcome: Percentage of Participants With ≥ 10 Points Improvement From Baseline in HRQoL Total Score at Months 1, 3, 6, 9, 12 and EoT
Description: as for outcome 27
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 281 | 286 | 1132
  Month 1 | 46.6 | 53.8 | 57.0
  Month 3: number analyzed (Participants) | 278 | 286 | 1137
  Month 3 | 53.6 | 59.4 | 64.6
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | 56.9 | 62.9 | 66.1
  Month 9: number analyzed (Participants) | 261 | 264 | 1077
  Month 9 | 57.1 | 62.9 | 67.7
  Month 12: number analyzed (Participants) | 250 | 255 | 1049
  Month 12 | 58.4 | 62.4 | 69.0
  EoT: number analyzed (Participants) | 290 | 294 | 1163
  EoT | 56.2 | 61.6 | 68.4
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 46, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.36 to 2.43]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 46, analysis 1]; Test type: Superiority; p = 0.014, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.08 to 1.92]

48. Secondary Outcome: Percentage of Participants With 50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours at Months 1, 3, 6, 9, 12 and EoT
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to each visit.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 291 | 288 | 1158
  Month 1 | 46.7 | 55.2 | 62.0
  Month 3: number analyzed (Participants) | 282 | 288 | 1137
  Month 3 | 58.2 | 67.0 | 73.3
  Month 6: number analyzed (Participants) | 266 | 273 | 1107
  Month 6 | 63.2 | 71.8 | 76.6
  Month 9: number analyzed (Participants) | 264 | 261 | 1070
  Month 9 | 67.0 | 73.6 | 77.8
  Month 12: number analyzed (Participants) | 258 | 256 | 1048
  Month 12 | 72.9 | 75.4 | 81.3
  EoT: number analyzed (Participants) | 301 | 297 | 1184
  EoT | 69.1 | 73.1 | 79.5
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio was from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of incontinence episodes per 24 hours as a covariate; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [1.34 to 2.41]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio wa from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of incontinence episodes per 24 hours as a covariate; Test type: Superiority; p = 0.019, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.06 to 1.95]

49. Secondary Outcome: Percentage of Participants With Zero Incontinence Episodes Per 24 Hours Using the Last 7 Diary Days at Months 1, 3, 6, 9, 12 and EoT
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The percentage of participants with no incontinence episodes recorded during the 7-day micturition diary is reported.
Time Frame: Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 291 | 288 | 1158
  Month 1 | 17.2 | 26.4 | 27.9
  Month 3: number analyzed (Participants) | 282 | 288 | 1137
  Month 3 | 27.0 | 35.1 | 40.0
  Month 6: number analyzed (Participants) | 266 | 273 | 1107
  Month 6 | 32.3 | 39.9 | 44.7
  Month 9: number analyzed (Participants) | 264 | 261 | 1070
  Month 9 | 37.1 | 43.7 | 46.9
  Month 12: number analyzed (Participants) | 258 | 256 | 1048
  Month 12 | 41.9 | 47.3 | 52.5
  EoT: number analyzed (Participants) | 301 | 297 | 1184
  EoT | 38.9 | 45.1 | 49.7
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 48, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.26 to 2.19]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 48, analysis 1]; Test type: Superiority; p = 0.133, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.94 to 1.62]

50. Secondary Outcome: Percentage of Participants With Micturition Frequency Normalization at Months 1, 3, 6, 9, 12 and EoT
Description: The percentage of participants with micturition frequency normalization was defined as participants who had ≥ 8 micturitions/24 hours at baseline and < 8 micturitions/24 hours postbaseline at months 1, 3, 6, 9, 12 and EoT.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS with data available at each time point. Participants with less < 8 micturitions per 24 hours at baseline were not included in the analysis. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 290 | 287 | 1155
  Month 1 | 34.5 | 29.3 | 36.8
  Month 3: number analyzed (Participants) | 281 | 287 | 1135
  Month 3 | 36.7 | 36.6 | 46.6
  Month 6: number analyzed (Participants) | 265 | 272 | 1105
  Month 6 | 42.3 | 43.4 | 51.4
  Month 9: number analyzed (Participants) | 263 | 260 | 1069
  Month 9 | 44.5 | 41.9 | 52.5
  Month 12: number analyzed (Participants) | 257 | 255 | 1047
  Month 12 | 46.3 | 44.7 | 56.4
  EoT: number analyzed (Participants) | 300 | 296 | 1181
  EoT | 46.0 | 46.3 | 55.9
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio was from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of micturitions per 24 hours as a covariate; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.18 to 2.03]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 50, analysis 1]; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.12 to 1.95]

51. Secondary Outcome: Percentage of Participants With ≥ 1 Point Improvement From Baseline in PPBC at Months 1, 3, 6, 9, 12 and EoT
Description: as for outcome 33
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 281 | 287 | 1133
  Month 1 | 53.0 | 59.2 | 64.1
  Month 3: number analyzed (Participants) | 278 | 286 | 1137
  Month 3 | 61.9 | 65.7 | 72.5
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | 64.6 | 68.8 | 73.8
  Month 9: number analyzed (Participants) | 261 | 264 | 1077
  Month 9 | 65.5 | 68.9 | 75.1
  Month 12: number analyzed (Participants) | 251 | 255 | 1049
  Month 12 | 69.7 | 73.7 | 76.9
  EoT: number analyzed (Participants) | 290 | 294 | 1163
  EoT | 66.2 | 71.4 | 76.0
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio is from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline PPBC as a covariate; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.24 to 2.29]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio was from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline PPBC as a covariate; Test type: Superiority; p = 0.109, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.94 to 1.77]

52. Secondary Outcome: Percentage of Participants With Major (≥ 2 Points) Improvement From Baseline in PPBC at Months 1, 3, 6, 9, 12 and EoT
Description: as for outcome 33
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 281 | 287 | 1133
  Month 1 | 24.9 | 28.2 | 30.7
  Month 3: number analyzed (Participants) | 278 | 286 | 1137
  Month 3 | 31.3 | 33.9 | 42.8
  Month 6: number analyzed (Participants) | 260 | 272 | 1108
  Month 6 | 35.0 | 38.2 | 45.4
  Month 9: number analyzed (Participants) | 261 | 264 | 1077
  Month 9 | 37.5 | 40.9 | 47.0
  Month 12: number analyzed (Participants) | 251 | 255 | 1049
  Month 12 | 40.6 | 40.4 | 51.9
  EoT: number analyzed (Participants) | 290 | 294 | 1163
  EoT | 38.3 | 39.8 | 50.3
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 51, analysis 2]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.26 to 2.25]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 51, analysis 2]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.62, 95% CI 2-sided [1.22 to 2.16]

53. Secondary Outcome: Percentage of Participants Who Were Double Responders (≥ 50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours and at Least 10 Points Improvement on OAB-q Symptom Bother Scale) at Months 1, 3, 6, 9, 12 and EoT
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to each visit. The OAB-q is a self-reported questionnaire with items relating to symptom bother and HRQoL. The symptom bother portion consists of 8 items, rated on a 6-point Likert scale (1 through 6). The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 (least severity) to 100 (worst severity). A negative change from baseline indicated an improvement.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 274 | 279 | 1115
  Month 1 | 36.1 | 46.6 | 52.6
  Month 3: number analyzed (Participants) | 270 | 281 | 1109
  Month 3 | 47.8 | 55.5 | 65.1
  Month 6: number analyzed (Participants) | 250 | 267 | 1080
  Month 6 | 50.4 | 56.9 | 65.8
  Month 9: number analyzed (Participants) | 254 | 252 | 1048
  Month 9 | 53.1 | 61.9 | 69.2
  Month 12: number analyzed (Participants) | 245 | 248 | 1018
  Month 12 | 59.2 | 60.9 | 73.2
  EoT: number analyzed (Participants) | 289 | 292 | 1156
  EoT | 55.7 | 58.2 | 70.8
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio was from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of incontinence episodes per 24 hours and baseline OAB-q symptom bother scale as covariates; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.99, 95% CI 2-sided [1.50 to 2.62]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio is from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of incontinence episodes per 24 hours and baseline OAB-q symptom bother scale as covariates; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.35 to 2.36]

54. Secondary Outcome: Percentage of Participants Who Were Double Responders (≥ 50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours and at Least 10 Points Improvement on OAB-q HRQL Total Score) at Months 1, 3, 6, 9, 12 and EoT
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to each visit. The OAB-q is a self-reported questionnaire with items relating to symptom bother and HRQoL. The HRQoL portion consists of 25 HRQoL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each item was scored 1-6. The total score was calculated by adding the 4 HRQoL subscale scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 274 | 279 | 1115
  Month 1 | 28.5 | 36.6 | 40.9
  Month 3: number analyzed (Participants) | 270 | 281 | 1109
  Month 3 | 39.6 | 43.8 | 52.3
  Month 6: number analyzed (Participants) | 250 | 267 | 1080
  Month 6 | 41.6 | 47.9 | 55.3
  Month 9: number analyzed (Participants) | 254 | 252 | 1048
  Month 9 | 43.7 | 51.2 | 57.6
  Month 12: number analyzed (Participants) | 245 | 248 | 1018
  Month 12 | 46.9 | 50.4 | 60.6
  EoT: number analyzed (Participants) | 289 | 292 | 1156
  EoT | 44.3 | 49.0 | 59.2
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio was from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of incontinence episodes per 24 hours and baseline OAB-q HRQL total score as covariates; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.46 to 2.54]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 54, analysis 1]; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.20 to 2.09]

55. Secondary Outcome: Percentage of Participants Who Were Double Responders (≥ 50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours and at Least 1 Point Improvement on PPBC) at Months 1, 3, 6, 9, 12 and EoT
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to each visit. The PPBC is a validated, global assessment tool using a 6-point Likert scale on which participants rated their subjective impression of their current bladder condition. Participants assessed their bladder condition using this scale: 1. Does not cause me any problems at all; 2. Causes me some very minor problems; 3. Causes me some minor problems; 4. Causes me (some) moderate problems; 5. Causes me severe problems; 6. Causes me many severe problems.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 274 | 280 | 1116
  Month 1 | 32.1 | 37.1 | 46.0
  Month 3: number analyzed (Participants) | 270 | 281 | 1109
  Month 3 | 43.3 | 47.7 | 57.6
  Month 6: number analyzed (Participants) | 250 | 267 | 1080
  Month 6 | 46.8 | 52.1 | 60.6
  Month 9: number analyzed (Participants) | 254 | 252 | 1048
  Month 9 | 49.6 | 53.2 | 63.0
  Month 12: number analyzed (Participants) | 245 | 248 | 1018
  Month 12 | 57.6 | 60.1 | 67.0
  EoT: number analyzed (Participants) | 289 | 292 | 1156
  EoT | 52.9 | 57.5 | 65.1
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio was from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of incontinence episodes per 24 hours and baseline PPBC as covariates; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.28 to 2.26]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 55, analysis 1]; Test type: Superiority; p = 0.019, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.06 to 1.86]

56. Secondary Outcome: Percentage of Participants Who Were Triple Responders (≥ 50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours, ≥ 10 Points Improvement on OAB-q Symptom Bother Scale and ≥1 Point Improvement on PPBC) at Months 1, 3, 6, 9, 12 and EoT
Description: The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to each visit. The symptom bother portion of the OAB-q consists of 8 items, rated on a 6-point Likert scale (1 through 6). The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 (least severity) to 100 (worst severity). A negative change from baseline indicated an improvement.The PPBC is a validated, global assessment tool using a 6-point Likert scale on which participants rated their subjective impression of their current bladder condition. Participants assessed their bladder condition using this scale: 1. Does not cause me any problems at all; 2. Causes me some very minor problems; 3. Causes me some minor problems; 4. Causes me (some) moderate problems; 5. Causes me severe problems; 6. Causes me many severe problems.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 274 | 279 | 1115
  Month 1 | 29.9 | 35.5 | 42.8
  Month 3: number analyzed (Participants) | 270 | 281 | 1109
  Month 3 | 38.9 | 44.8 | 54.1
  Month 6: number analyzed (Participants) | 250 | 267 | 1080
  Month 6 | 42.4 | 46.1 | 55.9
  Month 9: number analyzed (Participants) | 254 | 252 | 1048
  Month 9 | 46.5 | 50.8 | 59.2
  Month 12: number analyzed (Participants) | 245 | 248 | 1018
  Month 12 | 51.4 | 53.6 | 63.7
  EoT: number analyzed (Participants) | 289 | 292 | 1156
  EoT | 47.4 | 51.4 | 61.7
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio was from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of incontinence episodes per 24 hours, baseline OAB-q symptom bother scale and baseline PPBC as covariates; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.40 to 2.46]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 56, analysis 1]; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 1.58, 95% CI 2-sided [1.19 to 2.09]

57. Secondary Outcome: Participants Who Were Triple Responders (≥ 50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours, ≥ 10 Points Improvement on OAB-q HRQL Total Score and ≥ 1 Point Improvement on PPBC) at Months 1, 3, 6, 9, 12 and EoT
Description: The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in a micturition diary for 7 days prior to each visit. The HRQoL portion of the OAB-q consists of 25 HRQoL items comprising 4 HRQoL subscales, each item was scored 1-6. The total score was calculated by adding the 4 HRQoL subscale scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.The PPBC is a validated, global assessment tool using a 6-point Likert scale on which participants rated their subjective impression of their current bladder condition. Participants assessed their bladder condition using this scale: 1. Does not cause me any problems at all; 2. Causes me some very minor problems; 3. Causes me some minor problems; 4. Causes me (some) moderate problems; 5. Causes me severe problems; 6. Causes me many severe problems.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: FAS population with data available at each time point. LOCF was used for EoT.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 302 | 299 | 1193
percentage of participants
  Month 1: number analyzed (Participants) | 274 | 279 | 1115
  Month 1 | 25.2 | 29.0 | 35.5
  Month 3: number analyzed (Participants) | 270 | 281 | 1109
  Month 3 | 33.3 | 39.1 | 45.9
  Month 6: number analyzed (Participants) | 250 | 267 | 1080
  Month 6 | 36.8 | 41.2 | 49.6
  Month 9: number analyzed (Participants) | 254 | 252 | 1048
  Month 9 | 39.0 | 44.0 | 51.3
  Month 12: number analyzed (Participants) | 245 | 248 | 1018
  Month 12 | 44.1 | 47.6 | 54.6
  EoT: number analyzed (Participants) | 289 | 292 | 1156
  EoT | 40.1 | 45.2 | 53.3
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg + Mirabegron 50 mg; Odds ratio was from a logistic regression model including treatment group, sex, age group (< 65, ≥ 65 years), previous study history and geographic region as factors and baseline mean number of incontinence episodes per 24 hours, baseline OAB-q HRQL total score and baseline PPBC as covariates; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.33 to 2.34]
Statistical Analysis 2: Comparison: Solifenacin 5 mg vs Solifenacin 5 mg + Mirabegron 50 mg; [analysis description as in outcome 57, analysis 1]; Test type: Superiority; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.08 to 1.89]

58. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and EoT in Postvoid Residual (PVR) Volume
Description: PVR volume was assessed by ultrasonography or a bladder scanner.
Time Frame: Baseline and Months 1, 3, 6, 9, 12
Population: SAF population with data available at each time point. LOCF was used for EoT.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 305 | 303 | 1206
mL
  Month 1: number analyzed (Participants) | 295 | 298 | 1170
  Month 1 | 3.179 (27.491) | 4.549 (33.973) | 7.894 (38.369)
  Month 3: number analyzed (Participants) | 293 | 292 | 1175
  Month 3 | 4.686 (29.354) | 3.233 (32.679) | 7.033 (37.328)
  Month 6: number analyzed (Participants) | 280 | 282 | 1144
  Month 6 | 1.596 (29.399) | 3.418 (31.864) | 6.708 (35.881)
  Month 9: number analyzed (Participants) | 272 | 268 | 1111
  Month 9 | 3.074 (32.897) | 3.436 (32.170) | 8.229 (40.313)
  Month 12: number analyzed (Participants) | 263 | 266 | 1084
  Month 12 | 2.002 (32.453) | 4.818 (33.764) | 7.946 (38.118)
  EoT: number analyzed (Participants) | 300 | 302 | 1194
  EoT | 1.747 (32.400) | 7.382 (42.916) | 8.522 (39.501)

ADVERSE EVENTS:
Time Frame: From first dose of double-blind study drug up to 30 days after last dose of double-blind study drug (up to 56 weeks)
Description: The total number of deaths data includes deaths reported after the abovementioned timeframe.
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Solifenacin 5 mg + Mirabegron 50 mg
All-Cause Mortality (participants affected / at risk) | 1/305 | 0/303 | 1/1206
Serious Adverse Events (participants affected / at risk) | 8/305 | 8/303 | 51/1206
Other Adverse Events (participants affected / at risk) | 27/305 | 33/303 | 115/1206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirabegron 50 mg (N=305) | Solifenacin 5 mg (N=303) | Solifenacin 5 mg + Mirabegron 50 mg (N=1206)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Enterocele (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2
Appendicitis (Infections and infestations) | 1 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0
Haematoma infection (Infections and infestations) | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 2
Superinfection bacterial (Infections and infestations) | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Long thoracic nerve palsy (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Hysterocele (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Appendicectomy (Surgical and medical procedures) | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 2
Colon polypectomy (Surgical and medical procedures) | 0 | 0 | 1
Cystocele repair (Surgical and medical procedures) | 1 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 0 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 0 | 1
Spinal operation (Surgical and medical procedures) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mirabegron 50 mg (N=305) | Solifenacin 5 mg (N=303) | Solifenacin 5 mg + Mirabegron 50 mg (N=1206)
Dry mouth (Gastrointestinal disorders) | 12 | 18 | 74
Nasopharyngitis (Infections and infestations) | 16 | 15 | 43

LIMITATIONS AND CAVEATS:
Due to lack of data integrity, one site's data were not included in the efficacy and safety analysis, and another site's data for 5 patients were not included in the efficacy analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.